

# STATISTICAL ANALYSIS PLAN

An integrated Phase I/IIa, randomized, double-blind, placebo controlled study to evaluate the safety, tolerability and pharmacokinetics of single and multiple ascending dose(s) of oral RP3128 (CRAC channel modulators) in healthy volunteers and to evaluate the effect on Late Phase Asthmatic Response(LAR) to allergen challenge in patients with mild asthma

### **Protocol Number:**

Inflamax Protocol Number: 15-MR-001

Final Version 2 – 22 March 2017

# **Clinical Research Organization:**

Inflamax Research Limited

1310 Fewster Drive

Mississauga, ON L4W 1A4 Canada

### **Sponsor:**

Rhizen Pharmaceuticals SA

Fritz-Courvoisier 40,

Ch-2300 La Chaux-de-Fonds,

Switzerland

22June2017

Final Version 1.0



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# STATISTICAL ANALYSIS PLAN Final Version Approvals

An integrated Phase I/IIa, randomized, double-blind, placebo controlled study to evaluate the safety, tolerability and pharmacokinetics of single and multiple ascending dose(s) of oral RP3128 (CRAC channel modulators) in healthy volunteers and to evaluate the effect on Late Phase Asthmatic Response(LAR) to allergen challenge in patients with mild asthma

| Written By: Signature: | , |
|------------------------------------------|---------------------|
| Tian Fang | Date: >> Jun 201 |
| Biostatistics, Inflamax Research Limited | |
| Reviewed By: | 00 % 0012 |
| Signature: | Date: 23 June 2017. |
| Prajak Barde | |
| Medical Director | |
| Rhizen Pharmaceuticals SA | |



Study: Study 15-MR-001

# **Revision History**

| VERSI | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|---|---|---|---|
| Draft 0.1 | 02FEB2017 | Draft 0.1 | |
| Draft 0.2 | 02JUN2017 | Revised per internal and external comments | Tian Fang |
| Draft 0.3 | 16JUN2017 | Revised per internal and external comments | David Yu, Tian<br>Fang |
| Final 1.0 | 22JUN2017 | Final 1.0 | |



Study: Study 15-MR-001

# TABLE OF CONTENTS

| 1 | GLOSSARY OF ABBREVIATIONS | 9 |
|---|---|---|
| 2 | INTRODUCTION | 11 |
| 3 | TUDY OBJECTIVES | 12 |
| 3.1 | Primary Objective | 12 |
| 3.2 | Secondary Objective | 12 |
| 3.3 | Brief Description | 12 |
| 3.4 | Subject Selection | 13 |
| 3.5 | Determination of Sample Size | 13 |
| 3.6 | Treatment Assignment | 13 |
| 3.7 | Administration of Study Medication | 14 |
| 4 | ENDPOINTS | 15 |
| 4.1 | Primary Endpoints | 15 |
| 4.2 | Secondary Endpoints | 15 |
| 5 | ANALYSIS POPULATION | 17 |
| 5.1 | Randomized Population | 17 |
| 5.2 | Safety Population | 17 |
| 5.3 | Pharmacokinetic (PK) Population | 17 |
| 5.4 | Protocol Deviations | 17 |
| 6 | GENERAL ASPECTS FOR STATISTICAL ANALYSIS | 18 |
| <b>6.1</b> 6. | Summary Statistics | 18 |
| 6.2 | Key Definitions | 19 |
| 6.3 | Attribution of Treatment-Emergent AE for Imcompleted AE date/time | 19 |



Sponsor: Rhizen Pharmaceuticals SA

| | EMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND CATION | 21 |
|----------------|--------------------------------------------------------|----|
| 7.1 Su | ubject Disposition and Withdrawals | 21 |
| 7.2 Ba | aseline Characteristics | 21 |
| 7.3 Tr | reatment Compliance | 22 |
| 8 <b>A</b> l | NALYSIS OF PHARMACOKINETICS | 23 |
| 8.1 M | easurements | 23 |
| 8.2 Co | ollection Schedule | 23 |
| | erived Data and Handling of Missing or below LLOQ data | |
| 8.3.1<br>8.3.2 | Derivation of PK Parameters | |
| 8.4 Da | ata Summarization | 25 |
| | ata Presentation | |
| | AFETY | |
| 9.1 Ad | dverse Events | 27 |
| 9.2 La | aboratory Evaluations | 28 |
| 9.2.1 | Collection Schedule | 28 |
| 9.2.2 | Derived and Imputed Data | |
| 9.2.3 | Data Summarization and Presentation | 30 |
| 9.3 Vi | ital Signs | 30 |
| 9.3.1 | Measurements | 30 |
| 9.3.2 | | |
| 9.3.3 | Derived and Imputed Data. | |
| 9.3.4 | Data Summarization and Presentation | 32 |
| 9.4 EC | CG | 32 |
| 9.5 Ph | nysical Examination | 33 |
| 9.6 Ca | ognitive Test | 34 |
| 10 | EXPLORATORY ANALYSES | 35 |
| 4.4 | INTERIM ANALYCEC | |
| 11 | INTERIM ANALYSES | |



| 12 | CHANGES TO PLANNED ANALYSES | 37 |
|---|---|---|
| 13 | APPENDIX: | 38 |
| APPEN | IDIX A LIST OF CLINICAL LABORATORY TESTS (PART 1-3) | 38 |
| APPEN | DIX B: PART 1 (SAD) – Schedule of Events | 39 |
| APPEN | IDIX C: PART 2 (MAD) — Schedule of Events | 41 |
| 14 | TABLE AND LISTING | 44 |
| Table 1 | 4.1.1.S/M Disposition of Subjects (SAD/MAD) Randomized Population | 45 |
| Table 1 | 4.1.2.S/M Summary of Demographics (SAD/MAD) Safety Population | 46 |
| Table 14 | 4.2.1.1.X.S RP3128 Plasma Concentrations (ng/mL) by Time Point (SAD) Safety Population < Dose | 48 |
| | 4.2.1.1.1.X.M RP3128 Plasma Concentrations (ng/mL) by Time Point (MAD) – Day 1 Safety tion <dose level=""></dose> | 49 |
| | 4.2.1.1.2.X.M RP3128 Plasma Concentrations (ng/mL) by Time Point (MAD) – Day 7 Safety tion <dose level=""></dose> | 50 |
| Table 1 | 4.2.1.2.X.S RP3128 – Summary of PK Parameters (SAD) PK Population <dose level=""></dose> | 51 |
| Table 1 | 4.2.1.2.1.X.M RP3128 – Summary of PK parameters (MAD) – Day 1 PK Population <dose level=""></dose> | 52 |
| Table 1 | 4.2.1.2.2.X.M RP3128 – Summary of C <sub>trough</sub> (MAD) PK Population <dose level=""></dose> | 53 |
| Table 1 | 4.2.1.2.3.X.M RP3128 – Summary of PK parameters (MAD) – Day 7 PK Population <dose level=""></dose> | 54 |
| Table 1 | 4.2.2.X.1.M Summary of Cytokines <expression value="">: Change from Baseline (MAD)</expression> | 55 |
| | 4.2.2.X.2.M ANCOVA Results of Cytokine <expression value=""> Change from Baseline to Day 7 (Prest-dose)/ Difference between Pre-dose and Post-dose on Day 7 (MAD)</expression> | |
| | 4.3.1.1.S/M Treatment-Emergent Adverse Events – Overall Summary (SAD/MAD) Safety tion | 57 |
| | 4.3.1.2.S/M Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (AD) Safety Population | 58 |
| | 4.3.1.3.S/M Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and um Intensity (SAD/MAD) Safety Population | 59 |
| | 4.3.1.4.S/M Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and um Relationship (SAD/MAD) Safety Population | 60 |



| Table 14.3.3.1.X.S/M Summary of <laboratory panel=""> (SAD/MAD)</laboratory> | . 61 |
|---|---|
| Table 14.3.3.2.X.S/M <laboratory panel="">: Shift Table from Baseline to End of Treatment Results (SAD/MAD) Safety Population</laboratory> | . 63 |
| Table 14.3.4.X.S/M Summary of Vital Signs Data by Treatment, Visit and Time Point (SAD/MAD) Safety Population | . 64 |
| Table 14.3.4.6.S/M Summary of Weight Data by Treatment and Time Point (SAD/MAD) Safety Population | ı <b>65</b> |
| Table 14.3.5.1.S/M Summary of Overall ECG Interpretation (SAD/MAD) Safety Population | . 66 |
| Table 14.3.5.X.S/M Summary of ECG Continuous Data (SAD/MAD) Safety Population | 67 |
| Table 14.3.6.1.S/M Summary of Mini-Mental State Examination (SAD/MAD) Safety Population | . 68 |
| Listing 16.1.7.S/M Randomization Scheme and Code (SAD/MAD) Randomized Population | . 69 |
| Listing 16.2.1.S/M Subject Disposition and Completion/Discontinuation (SAD/MAD) Randomized Population | . 70 |
| Listing 16.2.2.S/M Protocol Deviations (SAD/MAD) Safety Population | . 71 |
| Listing 16.2.3.S/M Exclusions from Analysis Populations (SAD/MAD) Randomized Population | . 72 |
| Listing 16.2.4.S/M Demographics and Informed Consent at Screening (SAD/MAD) Safety Population | . 73 |
| Listing 16.2.5.1.S/M Study Drug Administration and Compliance (SAD/MAD) Safety Population | .74 |
| Listing 16.2.5.2.S/M Pharmacokinetic Sample Collection Data (SAD/MAD) Safety Population | .75 |
| Listing 16.2.5.3.S Pharmacokinetic Parameters (SAD) PK Population | 76 |
| Listing 16.2.5.4.S/M Reasons Why Pharmacokinetic Parameters Could Not be Determined (SAD/MAD) | . 77 |
| Listing 16.2.6.1: Cytokine assessment | . 78 |
| Listing 16.2.7.1.S/M Adverse Events (SAD/MAD) Safety Population | .79 |
| Listing 16.2.7.2.S/M Deaths, Other Serious and Significant Adverse Events Safety Population (SAD/MAD). | . 80 |
| Listing 16.2.8.X.S/M <laboratory panel=""> (SAD/MAD) Safety Population</laboratory> | . 81 |
| Listing 16.2.8.X.S/M <laboratory panel="">: Abnormal Results (SAD/MAD) Safety Population</laboratory> | . 81 |
| Listing 16.2.8.7.S/M Viral Screen and TB Test at Screening (SAD/MAD) Safety Population | . 83 |
| Listing 16.2.8.8.S/M Drug and Alcohol Screen (SAD/MAD) Safety Population | .84 |
| Listing 16.2.9.1.S/M Vital Signs (SAD/MAD) Safety Population | . 85 |



| Listing 16.2.10.1.S/M Electrocardiogram (ECG) (SAD/MAD) Safety Population | 86 |
|---|---|
| Listing 16.2.10.2.S/M ECG: Abnormal Results – Listing (SAD/MAD) Safety Population | 87 |
| Listing 16.2.11.S/M Mini-Mental State Examination (SAD/MAD) Safety Population | . 88 |
| Listing 16.2.12.S/M Medical History (SAD/MAD) Safety Population | 89 |
| Listing 16.2.13.S/M Clinical Events (SAD/MAD) Safety Population | 90 |
| Listing 16.2.14.S/M Prior and Concomitant Medications (SAD/MAD) Safety Population | 91 |
| Listing 16.2.15.M Electroencephalogram at Screening (MAD) Safety Population | 92 |
| Figure 14.4.1.S/M – Mean Plasma RP3128 Concentrations – Linear Scale (SAD/MAD) | 93 |
| Figure 14.4.2.S/M – Mean Plasma RP3128 Concentrations – Semi-logarithmic Scale (SAD/MAD) | 94 |
| Figure 14.4.3.X.S/M–Individual Plasma RP3128 Concentrations – Linear Scale (SAD/MAD) | 95 |
| Figure 14.4.4.X.S/M–Individual Plasma RP3128 Concentrations – Semi-logarithmic Scale (SAD/MAD) | 95 |



Study: Study 15-MR-001

# **GLOSSARY OF ABBREVIATIONS**

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ALP | Alkaline Phosphatase |
| ALT (SGOT) | Alanine Aminotransferase |
| ANC | Absolute Neutrophil Count |
| ANCOVA | Analysis of Covariance |
| AST (SGPT) | Aspartate Aminotransferase |
| AUC | Area Under the Curve |
| AUC <sub>0-t</sub> | Area Under the Plasma-Concentration Time Curve from Zero Up to the Last Measurable time point |
| AUC <sub>0-inf</sub> | Area Under the Curve from Zero extrapolated to infinite time |
| BUN | Blood Urea Nitrogen |
| bpm | Beats per minute |
| CFB | Change from Baseline |
| CK | Creatinine kinase |
| CM | Concomitant Medication |
| Cav | Average concentration during the dosing interval |
| $C_{max}$ | Peak Drug Concentration |
| C <sub>min</sub> | Lowest observed plasma concentration in the dosing interval |
| Ctrough | Plasma concentration at the end of the dosing interval |
| CRAC | Calcium Release Activated Calcium Channel |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| FSH | Follicular Stimulating Hormone |
| GGT | Gamma Glutamyl Transpeptidase |
| HCV | Hepatitis C Virus |
| HIV | Human Immune Deficiency Virus |
| Hr | Hour |
| HV | Healthy Volunteers |



Sponsor: Rhizen Pharmaceuticals SA

| Abbreviation | Description |
|---|---|
| ICH | International Conference on Harmonization |
| IMP | Investigational Medicinal Product |
| LAR | Late Phase Asthmatic Response |
| LPS | Lipopolysaccharide |
| Kel | Apparent terminal elimination rate constant |
| MAD | Multiple ascending dose |
| MCH | Mean Corpuscular Hemoglobin |
| MCHC | Mean Corpuscular Hemoglobin Concentration |
| MCV | Mean Corpuscular Volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mmHg | Millimeters of mercury |
| MMSE | Mini Mental State Examination |
| MTD | Maximum Tolerated Dose |
| PCP | Phencyclidine |
| PFT | Pulmonary Function Test |
| PI | Principal Investigator |
| PK | Pharmacokinetic |
| PR | P wave, R wave interval |
| PT | Preferred Term |
| QRS | Q wave, R wave, and S wave complex |
| QTcB | QT wave complex corrected for heart rate using Bazette's formula |
| SAD | Single ascending dose |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| SDTM | Study Data Tabulations Model |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| SRC | Safety Review Committee |
| t <sub>1/2</sub> | Half life |
| TEAE | Treatment Emergent AE |
| T <sub>max</sub> | Time of C <sub>max</sub> |
| K <sub>el</sub> | Terminal Rate Constant |



Study: Study 15-MR-001

# 2 INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide a thorough description of statistical methods and presentation of the study data to be used for the analysis of data generated from the Single Ascending Dose (SAD) part and the Multiple Ascending Dose (MAD) part of the clinical trial described in protocol: "An integrated Phase I/IIa, randomized, double-blind, placebo controlled study to evaluate the safety, tolerability and pharmacokinetics of single and multiple ascending dose(s) of oral RP3128 (CRAC channel modulators) in healthy volunteers and to evaluate the effect on Late Phase Asthmatic Response(LAR) to allergen challenge in patients with mild asthma."

This SAP is based on protocol RP3128-1601 Final Version 2 dated 22March2017. This document provides the detail statistical analysis plan for the SAD part and the MAD part of the protocol.

The SAP includes details of data handling procedures and statistical methodology. The SAP also provides the shells for the Tables, Listings, and Graphs (TLGs) to be delivered to Rhizen Pharmaceuticals SA, Inc.

The final statistical analysis will proceed in accordance with this SAP as approved by both Rhizen Pharmaceuticals SA and Inflamax Research Limited. Any deviation from this SAP will be documented in the final Clinical Study Report (CSR).

For this study, the Study Data Tabulation Model (SDTM) as well as the Analysis Data Model (ADaM) specifications will be prepared by Inflamax Research and provided to the Sponsor. SDTM Model 1.4 and SDTM Implementation Guide (SDTM IG) version 3.2 will be used ADaM Model 2.1 and ADaM Implementation Guide (ADaM IG) version 1.0 will be used. SDTM/ADaM datasets will be provided separately for SAD and MAD parts.

The following documents were also reviewed in preparation of this SAP:

- Electronic Case Report Form (eCRF) SAD Final Version 1.0 dated 31OCT2016
- Electronic Case Report Form (eCRF) MAD Final Version 1.0 dated 31OCT2016
- eCRF Completion Guidelines SAD&MAD Final v1.0 dated 31OCT2016
- Data Management Plan Final v1.0 dated
- Codelist Details dated 28OCT2016
- Safety Monitoring Committee charter, version 2.0, dated 21DEC2016



Study: Study 15-MR-001

# 3 TUDY OBJECTIVES

The study objectives related to the SAD and MAD portion of the trial are described below.

# 3.1 PRIMARY OBJECTIVE

- Part 1 (SAD) to investigate the safety and tolerability of single ascending oral doses of RP3128 in Healthy Volunteers (HV).
- Part 2 (MAD) to investigate the safety and tolerability of once a day multiple ascending oral doses of RP3128 at three dose levels (highest safe doses identified in SAD) in HV.

# 3.2 SECONDARY OBJECTIVE

- Part 1 (SAD) To characterize the pharmacokinetic (PK) profile of single ascending oral doses of RP3128 in HV.
- Part 2 (MAD) To characterize the multiple dose PK profile of oral RP3128 at steady state when administered once day, at three dose levels in HV.
- Part 2 (MAD) To evaluate ex-vivo effect of RP3128 on various biomarkers (Th1, Th2 and Th17 cytokines) following Lipopolysaccharide (LPS) or CD3/CD28 stimulation.

# 3.3 BRIEF DESCRIPTION

This is a phase I, single-center, double-blind, randomized, placebo-controlled study to evaluate the safety, tolerability, and PK of single or multiple ascending dose (SAD or MAD) of RP3128 in healthy volunteers.

There were 5 cohorts in SAD and 3 cohorts in MAD. In the first part of the study (Part 1, SAD), single dose of RP3128/placebo was administered on Day 1. In the second part (Part 2, MAD), multiple doses of RP3128/placebo were administered once a day from Day 1 to Day 7. In both SAD and MAD, the cohorts were dosed sequentially so that a minimum of 8 days was allowed between dose of previous cohort and the initiation of next cohort. Progression to the next higher dose occurred only after confirming safety, tolerability and PK of existing dose. In case of safety concern, additional subjects may be added to cohort for safety assessment as per the decision of Safety Review Committee (SRC).

In addition, sentinel design was applied. Within each cohort, 2 sentinel subjects was dosed first for safety assessment. Safety and tolerability data up to 24 hours was reviewed along with any observation up to 36 hours by the investigator prior to dosing the remaining subjects at that dose level. The remainder of the cohort was dosed sequentially at least 48 hours after confirming safety and tolerability of sentinel cohort.



Study: Study 15-MR-001

# 3.4 SUBJECT SELECTION

Healthy male subjects and female subjects of non-childbearing between the ages of 18 and 45 years were randomized at the study site.

All subjects must give written informed consent to be enrolled into the study Subjects were considered eligible to participate in this study if all inclusion criteria was satisfied and no exclusion criteria was met at screening. Please refer to the Protocol for detailed inclusion/exclusion criteria.

# 3.5 DETERMINATION OF SAMPLE SIZE

The sample size has been selected without performing a power calculation to provide descriptive information on the safety, tolerability, and PK following administration of RP3128. This trial enrolled up to 56 HV (32 in SAD and 24 in MAD). Number of subjects enrolled in this study is in line with standard phase I studies and is considered sufficient to provide descriptive information on the pharmacokinetics, safety and tolerability of RP3128 while minimizing exposure to humans. The actual number of dose cohorts will depend upon the emerging safety data.

# 3.6 TREATMENT ASSIGNMENT

Subjects who entered the treatment phase was assigned a unique 4-digit randomization number in the format of XYZZ to identify study part (X), cohort number (Y) and subject identifier (ZZ). The first 2 randomization numbers XY01 and XY02 in each cohort represents the sentinel subjects in Part number X and cohort number Y. For SAD and MAD parts, X is 1 and 2 respectively. For the SAD part, number Y is denoted by 1 to 5 for 5 cohorts, whereas for MAD part the number Y is denoted by 1 to 3 for 3 cohorts. Once any subject or randomization number is assigned, it cannot be reassigned to any other subject.

Allocation to treatment was based on a predetermined random order. Randomization to RP3128 or placebo took place for each cohort separately. The randomization lists were generated by an unblinded staff at Inflamax Research using the computer program Statistical Analysis System (SAS®) and managed according to the site's standard operating procedures (SOPs). Separate randomization ratios were used for study SAD Part and MAD Part as indicated in the tables below.



Study: Study 15-MR-001

# **Dose escalation cohorts for Part 1 (SAD)**

| Cohort | Dose level | n | Sentinel cohort | Remaining cohort | Total cohort |
|---|---|---|---|---|---|
| | | | RP3128: Placebo | RP3128: Placebo | RP3128: Placebo |
| S1 | 25 mg | 4 | 1:1 | 2:0* | 3:1 |
| S2 | 50 mg | 6 | 1:1 | 3:1 | 4:2 |
| S3 | 100 mg | 6 | 1:1 | 3:1 | 4:2 |
| S4 | 200 mg | 8 | 1:1 | 5:1 | 6:2 |
| S5 | 400 mg | 8 | 1:1 | 5:1 | 6:2 |

<sup>\*</sup>Single blind (subject)

# **Dose escalation cohorts for Part 2 (MAD)**

| Cohort | Dose level | N | Sentinel cohort | Remaining cohort | Total cohort |
|---|---|---|---|---|---|
| | | | RP3128: Placebo | RP3128: Placebo | RP3128: Placebo |
| M1 | 25 mg | 8 | 1:1 | 5:1 | 6:2 |
| M2 | 100 mg | 8 | 1:1 | 5:1 | 6:2 |
| M3 | 400 mg | 8 | 1:1 | 5:1 | 6:2 |

# 3.7 ADMINISTRATION OF STUDY MEDICATION

Depending on the cohort, specific dose/doses of RP3128/placebo was dispensed by pharmacy staff during the study. RP3128/placebo capsules was administered orally in the morning with approximately 240 mL (8 fluid ounces) of water at room temperature by the subject. For SAD part, the doses in 5 planned cohorts were 25 mg, 50 mg, 100 mg, 200 mg and 400 mg. For MAD part, the doses in 3 planned cohorts were determined to be 25mg, 100mg, and 400mg considering the safety and PK profile of RP3128 in SAD.



Study: Study 15-MR-001

# 4 ENDPOINTS

# 4.1 PRIMARY ENDPOINTS

The primary endpoints for both SAD and MAD parts are as follows:

- Incidence of AEs
- Changes in vital signs (blood pressure, pulse rate, respiratory rate, oral temperature) and weight
- Changes in 12-lead ECG parameters
- Changes in clinical laboratory assessments (hematology, chemistry, urinalysis)

# 4.2 SECONDARY ENDPOINTS

The secondary endpoints include PK parameters and biomarker assessments

# SAD-PK Endpoints:

- Maximum observed plasma concentration (C<sub>max</sub>)
- Time to maximum observed plasma concentration (T<sub>max</sub>)
- Area under the plasma concentration-time curve from time zero until the last time point with measurable concentration (AUC<sub>0-t</sub>)
- Area under the plasma concentration-time curve from time zero to infinity (AUC<sub>0-inf</sub>)
- Apparent termination elimination rate constant (K<sub>el</sub>)
- Apparent terminal elimination half-life  $(t_{1/2})$

# MAD-PK Endpoints:

- Maximum observed plasma concentration in the dosing interval  $(C_{max})$  (Day 1, Day 7)
- Lowest observed plasma concentration in the dosing interval (C<sub>min</sub>) (Day 7)
- Plasma concentration at the end of the dosing interval (C<sub>trough</sub>) (Day 3, Day 5, Day 7)
- Average concentration during the dosing interval (C<sub>av</sub>) (Day 7)
- Time to maximum plasma concentration (T<sub>max</sub>) (Day 1, Day 7)
- Area under the plasma concentration-time curve from time zero until the last time point with measurable concentration (AUC<sub>0-24</sub>) (Day 1, Day 7)
- Degree of fluctuation [(C<sub>max</sub>-C<sub>min</sub>)/C<sub>av</sub>] (Day 7)
- Swing  $[(C_{max}-C_{min})/C_{min}]$  (Day 7)
- Terminal half-life  $(t_{1/2})$  (Day 1, 7)



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# MAD-Biomarker Endpoints:

• Levels of various biomarkers (Th1, Th2 and Th17 cytokines) following LPS or CD3/CD28 stimulation



Study: Study 15-MR-001

# 5 ANALYSIS POPULATION

# 5.1 RANDOMIZED POPULATION

The randomized population consists of all eligible subjects who are randomized to receive a treatment regardless whether they are actually treated. These subjects are grouped by their randomized treatment group. The randomized population will be used to summarize subject disposition from randomization through termination.

# 5.2 SAFETY POPULATION

The Safety population will include randomized subjects who receive at least one dose of study drug (RP3128 or placebo) during treatment phase. Subjects will be analyzed as treated, if any subjects received the study drug different from the drug they were randomized to receive. There will be separate safety populations each for SAD and MAD parts. The Safety population will be used for all analyses of safety endpoints, biomarker endpoints, as well as demographics and baseline characteristics.

# 5.3 PHARMACOKINETIC (PK) POPULATION

The PK population will include all safety subjects with sufficient concentration-time data to determine PK parameters and no major protocol deviations. The PK population will be used for all analyses of PK endpoints.

# 5.4 PROTOCOL DEVIATIONS

All protocol deviations related to study inclusion or exclusion criteria, conduct of the trial, subject management or subject assessment will be listed. The list of protocol deviations will be reviewed by the Sponsor, the PI, the study statistician and the study scientist before unblinding the study.



Study: Study 15-MR-001

# 6 GENERAL ASPECTS FOR STATISTICAL ANALYSIS

# 6.1 SUMMARY STATISTICS

The standard summary statistics that will be calculated for quantitative and qualitative variables are:

# • Ouantitative:

- Standard Statistics for both Safety/PK: Number of subjects, mean, median, standard deviation (SD), minimum and maximum of the raw data
- Additional Statistics for PK: coefficient of variance (PK concentration and PK parameters), geometric mean, and geometric CV (%) ( PK parameters AUC and Cmax in SAD part and AUC<sub>0-24</sub>, C<sub>max</sub>, C<sub>min</sub>, C<sub>trough</sub> in MAD part)
- Qualitative: number of subjects (n), number of missing observations (nmiss), absolute and relative frequencies (%) per category.

Demographics and disposition will be summarized by treatment group and overall.

Data collected pre- and post-dose during the treatment period (e.g., vital signs, ECG, and clinical laboratory) will be summarized by treatment group (dose level), visit and/or time point. For quantitative variables (ECG measurements, vital signs, hematology, etc.), change from baseline will be calculated and summarized by treatment, visit and/or time point together with baseline and post-dose value. For qualitative variables (e.g., ECG interpretation, urinalysis), standard summary of frequencies will be calculated by treatment, visit and/or time points. For safety lab data only, shift table will be produced to present the change of reference range indicator from baseline to post-dose. PK parameters will be summarized by treatment group, and visit (if applicable). All subjects assigned and treated with Placebo in different cohorts will be pooled together and summarized as a single group.

# **6.1.1** Summary Statistics Reporting Precision

Summary statistics will be presented to the following degree of precision:

Table 1. Reporting Precision

| Statistics | Degree of Precision |
|---|---|
| Mean (of all kinds), Median | One more decimal place than the raw data |
| Standard deviation, Standard error | Two more decimal places than the raw data |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

| Minimum, Maximum | The same number of decimal places as the raw data |
|---|---|
| Percent, Coefficient of Variance | Two decimal places for PK parameters, and one decimal place for all other parameters |
| PK Concentration, AUC, Cmax | The same number of decimal places as LLOQ |

All fractional numeric values will be presented with a zero to the left of the decimal point (for example, 0.12, -0.30, not .12, -.30).

#### 6.2 **KEY DEFINITIONS**

The day of administration of the first dose of study drug during the treatment period is defined as Study Day 1. Study Day -1 is the day before dosing, all assessments prior to Study Day 1, including the Screening and Check-in Visits, will have negative study days.

The baseline observation will be the last non-missing value prior to the first dose of study drug.

Nominal Time is the scheduled measurement time relative to time 0. Time 0 is precisely defined for each analysis below.

For AEs, onset time from dosing will be calculated as the difference between the event and dosing start date/time. Onset time from dosing will be expressed in days, hours and minutes. If time is missing, onset time from dosing will be calculated as the difference between the start date and dosing date plus 1 and expressed in days when the event date is on or after the dosing date; otherwise, onset time from dosing will be calculated only as difference between the start date and dosing date and expressed in negative numbers.

Duration will be calculated for AEs that resolve as the difference between the AE resolution date/time and onset date/time and will be expressed in days, hours and minutes. If time is missing, duration will be calculated as the difference between the resolution date and onset date plus 1 and expressed in days. AE onset time from dosing and duration of AE will only be derived when both start and end dates are complete.

### 6.3 ATTRIBUTION OF TREATMENT-EMERGENT AE FOR **IMCOMPLETED AE DATE/TIME**

AEs with incomplete start dates and times will be attributed to treatment according to the following algorithm:

1. Only the year is reported: If the year is after the year of the dose, the event will be considered as treatment-emergent. If the year is the same as the day of the dose, the event will not be considered as treatment-emergent.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

2. Only the month and year are reported: If the month is after the month of the first dose, event will be considered as treatment-emergent. If the month is the same as the month of the first dose, the event will not be considered as treatment-emergent.

3. Only the time is missing: If the event occurred on or after the day of the first dose in the treatment period, then the event will be considered as treatment-emergent. Otherwise, the event will not be considered as treatment-emergent.



Study: Study 15-MR-001

# 7 DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION

# 7.1 SUBJECT DISPOSITION AND WITHDRAWALS

For subject disposition, the following frequencies (number and percent) will be displayed by treatment group and overall for the randomized population:

- Subjects in the Randomized Population (number only)
- Subjects in the Safety Population (number only)
- Subjects in PK population
- Subjects who completed the study
- Subjects who discontinued early, as well as reasons for subject discontinuation

The denominators for the percent calculations will be the number of safety subjects per treatment group or overall.

A listing of randomization scheme will include the subject's identification, cohort, date of randomization, and treatment assignment.

Subjects' completion/discontinuation status will be listed by cohort/treatment and will include date of completion/early discontinuation, date of dosing and, for those who discontinued early, the specific reason(s) for discontinuation.

All deviations captured in eCRF will be listed. The list of protocol deviations will be reviewed by the Sponsor, the PI, the lead statistician and the study scientist and finalized before unblinding the treatment.

A listing of subjects excluded from the analysis populations will also be produced.

# 7.2 BASELINE CHARACTERISTICS

Demographics (age, sex, race, ethnicity), informed consent date, weight, height and BMI at screening will be listed and summarized using descriptive statistics (number of subjects, mean, standard deviation, minimum, median and maximum for quantitative variables and the proportion of subjects for qualitative variables) by treatment group and overall for the safety population. No formal statistical comparison between groups will be performed.

Concomitant medication/medical history data, including clinical events, will be listed for all safety subjects.



Study: Study 15-MR-001

# 7.3 TREATMENT COMPLIANCE

Subject must take study drug at the study site. Failure of treatment compliance will lead to termination of study. The necessary measures will be employed to ensure treatment compliance. The study drug will be dispensed or administered according to applicable standard operating procedures (SOPs). Study drug administration will be listed and ordered by cohort, treatment, subject and visit/day.



Study: Study 15-MR-001

# 8 ANALYSIS OF PHARMACOKINETICS

The PK population will be used for all PK analysis and listings.

# 8.1 MEASUREMENTS

A 4 ml of blood sample were collected at each planned time point for measurement of drug concentration in plasma. The time and date of collection of each sample was recorded in CRF.

# 8.2 COLLECTION SCHEDULE

For SAD part, blood samples will be collected for plasma levels of RP3128 on Day 1 (Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0, 8.0, 12.0, 24.0 and 48 hr), Day 5, Day 8 and Day 15. For MAD part, blood samples will be collected for plasma levels of RP3128 on Day 1 (Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0, 8.0, 12.0 and 24.0 hr), Day 3, Day 5, Day 7 (Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0, 8.0, 12.0 and 24.0 hr), Day 9 (48 hr), Day 10 (72 hr), Day 11 (96 hr), Day 12 (120 hr), Day 13 (144 hr) and Day 15 (192 hr).

# 8.3 DERIVED DATA AND HANDLING OF MISSING OR BELOW LLOQ DATA

### **8.3.1** Derivation of PK Parameters

PK parameters for RP3128 will be derived with validated SAS programs for all RP3128 dose levels by non-compartmental analysis of the plasma concentration data using actual sampling times.

The following pharmacokinetic variables will be derived:

# SAD:

- Maximum observed plasma concentration (C<sub>max</sub>)
- Time to maximum plasma concentration (T<sub>max</sub>)
- Terminal half-life  $(t_{1/2})$
- Area under the plasma concentration-time curve from time zero until the last measurable time point (AUC<sub>0-t</sub>)
- Area under the plasma concentration-time curve from time zero to infinity time (AUC<sub>0-inf</sub>)
- Elimination rate constant (K<sub>el</sub>)

# MAD:

Maximum observed plasma concentration in the dosing interval (C<sub>max</sub>) (Day 1, Day 7)



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

- Lowest observed plasma concentration in the dosing interval (C<sub>min</sub>) (Day 7)
- Plasma concentration at the end of the dosing interval (C<sub>trough</sub>) (Day 3, Day 5, Day 7)
- Average concentration during the dosing interval (C<sub>av</sub>) (Day 7)
- Time to maximum plasma concentration (T<sub>max</sub>) (Day 1, Day 7)
- Area under the plasma concentration-time curve from time zero until the last time point with measurable concentration (AUC<sub>0-24</sub>) (Day 1, Day 7)
- Degree of fluctuation  $[(C_{max}-C_{min})/C_{av}]$  (Day 7)
- Swing  $[(C_{max}-C_{min})/C_{min}]$  (Day 7)

The PK parameters will be estimated as follows:

- The  $C_{max}$  and the corresponding  $T_{max}$ ,  $C_{min}$  and  $C_{trough}$  will be read directly from the concentration-time plot (observed data, not predicted data by the program).
- AUCs will be calculated using the linear trapezoidal rule.
- The terminal elimination rate constant (K<sub>el</sub>) will be determined by log linear regression obtained on at least the 3 last quantifiable concentrations and will not include C<sub>max</sub>. The adjusted square of the correlation coefficient (R-square adjusted) for the goodness of fit of the regression line through the data points must be at least 0.80 for the K<sub>el</sub> value to be considered reliable. If fewer than 3 quantifiable concentrations are available after Cmax or if R-square is less than 0.80, the K<sub>el</sub> will be left uncalculated.
- $t_{1/2}$  is calculated by the program as  $ln2/K_{el}$ . If  $K_{el}$  is not calculable, then  $t_{1/2}$  will also remain missing.
- The AUC from 0 to infinity is calculated by the program as:

  AUC<sub>0-inf</sub> = AUC<sub>0-t</sub> + AUC<sub>t-inf</sub> where t is the sampling time point of the last measurable concentration. AUC<sub>t-inf</sub> is calculated by the program as: C<sub>t</sub>/ K<sub>el</sub>, where C<sub>t</sub> is the observed concentration at time t and K<sub>el</sub> is the elimination rate constant during the apparent terminal elimination phase. If K<sub>el</sub> is not calculable, AUC<sub>0-inf</sub> will be set to missing.
- The AUC extrapolation to infinity (AUC<sub>t-inf</sub>) must be  $\leq$ 20% of the total area for AUC<sub>0-inf</sub> to be considered reliable.

# 8.3.2 Handling of Missing Plasma Concentration Data or below LOQ

Plasma concentrations can only be missing if the sample was not collected. These missing concentrations will be considered as non-informative missing and will not be imputed.

However, if a plasma sample was collected, but the resulting assay failed to detect a quantifiable concentration, these will be imputed in the following way:

• Concentration values below the assay's lower limit of quantification (<lower limit of quantification (LLOQ) or below the limit of quantification (BLQ)) in pre-dose samples and



RESEARCH Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

in samples taken before the time of the first quantifiable concentration will be treated as zero.

- All sample collected prior to dosing will be treated as zero.
- Post-dose BLQ values after the first quantifiable time point that are flanked and followed by quantifiable concentrations will be set to LLOQ.
- Post-dose BLQ values after the first quantifiable time point that are not followed by quantifiable concentrations will be set to LLOQ.
- For PK profiles with no values reported above the LLOQ, these BLQ values will be set to LLOQ.

# 8.4 DATA SUMMARIZATION

PK parameters and plasma concentration data will be summarized by treatment using the following descriptive statistics (Table 2):

Table 2. PK Summary Statistics

| Variable | Summarized with: |
|---|---|
| Plasma concentration at each time point | n, arithmetic mean, SD, CV%, minimum, median and maximum |
| AUCs, C <sub>max</sub> , C <sub>min</sub> , C <sub>trough</sub> , C <sub>av</sub> | n, arithmetic mean, SD, CV% (calculated as 100%*SD/mean), minimum, median, maximum, geometric mean and geometric CV% (calculated as $CV = 100\% \times \sqrt{e^{z^2} - 1}$ , where $z^2$ is the variance of $ln(PK)$ parameter) |
| t <sub>1/2</sub> , K <sub>el</sub> , T <sub>max</sub> ,degree of fluctuation, swing | n, arithmetic mean, SD, CV%, minimum, median, maximum |

Samples taken outside the sampling windows may be excluded from by-time point summary statistics; this will be determined prior to unblinding.

# 8.5 DATA PRESENTATION

The actual sampling time of PK blood sample collection will be listed for each cohort and will include the deviation in time from the protocol scheduled time, if applicable.

Individual subject plasma concentration data will be listed by subject, time point and treatment and will be summarized at each time point by treatment group for the Safety population. Individual subject PK parameters will be listed in a table by subject and will be summarized by treatment group for the PK population.



Study: Study 15-MR-001

PK parameters of secondary interest, namely R-square adjusted, the number of data points used for estimating  $K_{el}$ , the upper and lower time point used for estimation of  $K_{el}$ , and the % AUC extrapolation from  $t_{last}$  (last time point of blood draw) to infinity will be listed by subject and dose level/cohort to enable verification of the exclusions, if any, of data from the summary statistics of the PK parameters of primary interest.



Study: Study 15-MR-001

# 9 SAFETY

The analysis population used for safety analyses will be the Safety population. Safety will be assessed on the basis of AE, clinical laboratory data, vital signs, ECG parameters, MMSE and physical examinations.

# 9.1 ADVERSE EVENTS

All subjects in the Safety population will be included in the adverse event analysis.

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary (Version 19.1 or higher)

An AE is defined as any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom (for example, an abnormal laboratory finding), or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no study treatment has been administered.

In this study, all AEs that occur after any subject has been screened through the post-treatment follow-up period, whether or not they are related to the study, must be recorded on the eCRF, and must include the following: date and time of onset, date and time of resolution, severity, seriousness, causality (relationship to study medication), actions required, and outcome. Clinically significant and severe AEs must be examined to determine whether they meet criteria of a dose-limiting toxicity.

A treatment-emergent AE (TEAE) is any that is new in onset or was aggravated in severity or frequency following the first dose of study drug, up to and including the last visit of the study. Treatment emergence will be determined by comparing the AE start date/time with the actual date/time of first dose. In the case that the AE start date/time are incomplete, treatment emergence will be imputed according to the algorithm in SAP Section 6.5.

Adverse events will be listed chronologically by cohort/treatment, subject and AE start date/time. This listing will include all data collected in the eCRF, along with the derived variables: onset time since first dose, duration of AE and the coded variables system organ class (SOC) and preferred term (PT). Time since dose and duration will be calculated as described in SAP Section 6.3. In addition, serious AEs (SAEs) will be listed separately, if any occurs.

The summary of AEs will be limited to TEAEs only. In cases where severity is missing for a TEAE, the TEAE will be considered to be the highest degree of severity: Severe. In cases where relationship information is missing for a TEAE, the TEAE will be considered to be reasonably related. Displays of TEAEs will include:



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# • Overall Summary of TEAEs

This table will include the number of events, number and percent of subjects who experienced TEAEs, serious TEAEs, severe TEAEs, related TEAEs and TEAEs leading to study discontinuation, summarized by treatment group.

• Summary of TEAEs by SOC, PT and Treatment Group

A summary of the number of events, number and percent of subjects who experienced at least one TEAE, as well as the number of events, number and percent of subjects who experienced each specific SOC, and PT will be presented by treatment group (including pooled placebo and pooled RP3128). If a subject has more than one occurrence of the same PT then the PT will be counted only once for that subject under the SOC at which it was experienced.

• Summary of TEAEs by SOC, PT, Treatment Group and Maximum Severity

A summary of the number and percent of subjects who experienced at least one TEAE by maximum severity as well as the number and percent of subjects who experienced each specific SOC and PT by maximum severity will be presented by treatment group. For this analysis, if a subject has more than one occurrence of the same PT, then the PT will be counted only once for that subject under the maximum severity at which it was experienced.

• Summary of TEAEs by SOC, PT, Treatment Group and Maximum Relationship

A summary of the number and percent of subjects who experienced at least one TEAE by maximum relationship as well as the number and percent of subjects who experienced each specific SOC and PT by maximum relationship will be presented by treatment group. For this analysis, if a subject has more than one occurrence of the same PT, then the PT will be counted only once for that subject under the maximum relationship at which it was experienced.

# 9.2 LABORATORY EVALUATIONS

All subjects in the Safety population will be included in the safety laboratory analysis.

# 9.2.1 Collection Schedule

At screening, Serology, Tuberculin test / QuantiFeron- TB®-Gold test, Alcohol and urine drug screening will be done to assess eligibility for the study. Drug screening includes opiates, methadone, cocaine, amphetamine, cannabinoids, barbiturates, and benzodiazepines. Alcohol will be screened using alcohol breath test. If the subject has a positive result, the subject will be considered a screen failure and must be excluded from the study. The result will be listed by cohort/treatment, subject and visit.

Female subjects will undergo a serum pregnancy test (quantitative β-HCG) test at screening.



Study: Study 15-MR-001

UPT (Urine pregnancy tests) will be performed at later time points in case of suspected pregnancy. The result will be listed by cohort/treatment, subject and visit.

Follicular Stimulating Hormone (FSH) will be evaluated at screening to confirm postmenopausal status for the females who reported having no menses less than 12 months.

For SAD part, the clinical laboratory evaluations, including Clinical chemistry, hematology, serum electrolyte, coagulation and urinalysis, will be performed at screening, Day -1, Day 2, Day 3, Day 8 and Day 15. For MAD part, the clinical laboratory evaluations, including Clinical chemistry, hematology, serum electrolyte, coagulation and urinalysis, will be performed at screening, Day -1, Day 2, Day 5, Day 7, Day 8 and Day 15. If blood, nitrites or leukocytes are abnormal, automatically microscopic urinalysis will be performed. Additional investigations will be performed if clinically indicated.

Laboratory assessment times are shown below in Table 3.

Table 3. Laboratory Parameters Assessment Times

| Visit/Day | Clinical<br>Laboratory | Serology | FSH | Drug<br>and<br>alcohol<br>screen | Pregnancy testing |
|---|---|---|---|---|---|
| Screening | <b>✓</b> | ✓ | ✓ | ✓ | ✓ |
| Day -1<br>(Check-in) | <b>✓</b> | | | ✓ | <b>✓</b> |
| Day 2 | <b>✓</b> | | | | |
| Day 3 | ✓(SAD) | | | | |
| Day 5 | ✓(MAD) | | | | |
| Day 7 | ✓(MAD) | | | | |
| Day 8 | <b>✓</b> | | | | |
| Day 15 | <b>✓</b> | | | | |



Study: Study 15-MR-001

# 9.2.2 Derived and Imputed Data

Some numeric lab values may be reported as '>n.n' or <n.n; these will be analyzed in the summary statistics as n.n. For example, potassium recorded as >9.0 mmol/L would be summarized as 9.0 mmol/L.

Baseline is defined as the last non-missing observation prior to first dosing on Day 1.

# 9.2.3 Data Summarization and Presentation

Laboratory sample data and values from laboratory assessments will be listed chronologically by cohort/treatment, subject, and visit. Abnormal findings in laboratory data will be listed with a flag for clinical significance based on investigator judgment. Abnormal laboratory findings will also be provided in a separate listing.

For quantitative data, change-from-baseline (CFB) will be calculated as the difference between the post-dose visit and baseline. For the SAD part, CFB will be calculated for Day 2, Day 3 (at discharge), Day 8, and Day 15. For the MAD part, CFB will be calculated for Day 2, Day 5, Day 7, Day 8 (at discharge), and Day 15.

The laboratory will assign a reference range indicator to all test results by comparing the actual test value to the reference range. The quantitative results will have indicator values of Low, High, and Normal, while the qualitative results will have indicator values of Normal and Abnormal. The investigator or designee will review non-normal results to judge their clinical significance.

Quantitative results will be summarized for baseline, post-dose visits and CFB values by treatment group using standard summary statistics (n, mean, SD, minimum, median and maximum). Qualitative results (e.g., some tests in urinalysis) will be summarized by treatment group using frequency and percentage. The reference range indicator data will also be tabulated using frequency and percentage for both quantitative and qualitative results. No inferential tests will be conducted on lab data.

In addition, 3 by 3 shift tables will be produced to compare the change in reference range indicator from baseline to Day 3 for the SAD / Day 8 for the MAD part for each laboratory test. For parameters where only two possible values are available (i.e., Normal and Abnormal), the Abnormal values will be counted as High (H) in the 3 by 3 table.

# 9.3 VITAL SIGNS

All subjects in the Safety population will be included in the vital signs analysis.

# 9.3.1 Measurements

Vital signs will consist of blood pressure (systolic and diastolic blood pressure, mmHg), heart rate (beats per minute (bpm)), respiratory rate (breaths/min), temperature (°C) and weight. At

Page 30 of 95



Study: Study 15-MR-001

screening, vital signs will be assessed in the supine position after the subject has rested for at least 3 minutes. Blood pressure and pulse will be assessed again after three minutes in the standing position. At other time points, vitals will be measured after 3 minutes supine rest. Vitals should be completed within +/- 30 minute of schedule timing to avoid overlapping.

Height and weight (without shoes) will be collected at Screening and BMI will be calculated. Height, weight and BMI will be collected and calculated at other time points (check-in, follow-up and ET visit).

# 9.3.2 Collection Schedule

For SAD, vital signs on screening, Day -1 (at the time of admission), Day 1 (pre-dose, 30 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose), Day2, Day 3, Day 5, Day 8 and Day 15. For MAD, vital signs on screening, Day -1 (at the time of admission), Day 1 & Day 2 (pre-dose, 30 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose), Day 3, Day 4, Day 5, Day 6, Day 7 (pre-dose, 30 min, 1, 2, 4, 6, 12 hrs post dose), Day 8, Day 9, Day 11 and Day 15. Assessment times for vital sign parameters are presented below in Table 4 & 5.

**Table 4. Vital Sign Assessment Times (SAD)** 

| Visit/Day | Vital Sign Assessment Times |
|-------------------|----------------------------------------------------------|
| Screening | ✓ |
| Check-in Day -1 | ✓ |
| Day 1 (Treatment) | pre-dose, 30 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose |
| Day 3 (Discharge) | ✓ |
| Day 5 | ✓ |
| Day 8 | ✓ |
| Day 15 | ✓ |

Table 5. Vital Sign Assessment Times (MAD)

| Visit/Day | Vital Sign Assessment Times |
|-----------------|-----------------------------|
| Screening | ✓ |
| Check-in Day -1 | ✓ |



Study: Study 15-MR-001

| Day 1 (Treatment) | Pre-dose, 30 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose |
|-------------------|----------------------------------------------------------|
| Day 3 (Treatment) | ✓ |
| Day 4 (Treatment) | ✓ |
| Day 5 (Treatment) | ✓ |
| Day 6 (Treatment) | ✓ |
| Day 7 (Treatment) | Pre-dose, 30 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose |
| Day 8 (Discharge) | ✓ |
| Day 9 | ✓ |
| Day 11 | ✓ |
| Day 15 | ✓ |

# 9.3.3 Derived and Imputed Data

Baseline will be defined as the last non-missing observation prior to the dosing on Day 1.

# 9.3.4 Data Summarization and Presentation

Vital signs data will be listed chronologically by cohort/treatment, subject, visit/day, and time point when applicable.

Baseline values, absolute values and change from baseline for each post-dose time point will be summarized by treatment group using standard descriptive statistics. Off-treatment vital signs (e.g., Screening, Day -1, Unscheduled visit) will be listed but not otherwise analyzed. No inferential tests will be conducted.

Weight (without shoes) is measured at screening, check-in, follow-up and ET visit, the screening observation is used to summarize demographics, and the last non-missing observation prior to dosing on Day 1 (mostly likely the check-in observation) is defined as baseline to calculate weight change at post-doing visits.

# **9.4** ECG

All subjects in the Safety population will be included in the ECG analysis.

For SAD, a standard 12-lead ECG will be performed with the subject in a supine position at



Study: Study 15-MR-001

Screening, Day -1 (at the time of admission), Day 1 (pre-dose, 15, 30, 45 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose), Day 3, Day 5, Day 8 and Day 15 or Early Termination. For MAD, a standard 12-lead ECG will be performed with the subject in a supine position at Screening, Day -1 (at the time of admission), Day 1 (pre-dose, 15, 30, 45 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose), Day 5, Day 7 (pre-dose, 15, 30, 45 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose), Day 8 and Day 15 or Early Termination. Triplicate ECG will be taken 1 minute apart on screening, Day 1 (pre-dose) and for confirmation of abnormality detected in the single ECG measurement based on Investigator judgement.

For each assessment, the ECG will be reviewed by the qualified physician and the interpretation will be recorded in the eCRF as normal, abnormal but not clinically significant, abnormal and clinically significant. In addition, the standard ECG parameters including ventricular rate (VR), and intervals for PR, QRS, QT, and QTcB (Bazette's corrections for heart rate) will be recorded.

Baseline will be defined as the last non-missing observation prior to dosing on Day 1.

All ECG data will be listed chronologically by cohort/treatment, subject, visit/day, and time point. Abnormal ECG results will be provided in a separate listing.

Overall interpretation of ECG measurements will be summarized by treatment at each time point using frequencies. Baseline values, absolute values, and CFB will be summarized by treatment group using standard descriptive statistics for VR, PR interval, QRS duration, and QT interval. Off-treatment ECG data (e.g., Screening, Day -1, and Unscheduled visits) will be listed but not otherwise analyzed. No inferential tests will be conducted on ECG data.

# 9.5 PHYSICAL EXAMINATION

For SAD, a complete physical examination will be performed at screening, Day -1, Day 3, Day 8 and Day 15, or if necessary at the Early Termination visit. For MAD, a complete physical examination will be performed at screening, Day -1, Day 4, Day 8 and Day 15, or if necessary at the Early Termination visit. This exam will include general appearance, skin, neck (including thyroid), eyes, ears, nose, throat, lungs, heart, abdomen, back, lymph nodes, extremities, vascular, and neurological. If indicated based on medical history and/or symptoms, rectal, external genitalia, breast, and/or pelvic exams may be performed. Information for all physical examinations must be included in the source documentation at the study site and will not be recorded the CRF. Significant findings that are present prior to informed consent are included in the Relevant Medical History CRF. Significant findings observed after informed consent signature which meet the definition of an Adverse Event must be appropriately recorded on the Adverse Event CRF. No listings and summary tables will be produced separately.



Study: Study 15-MR-001

# 9.6 COGNITIVE TEST

A cognitive test (e.g. Mini-Mental State Examination (MMSE)) will be performed at Screening and Day 3 (SAD)/ Day 8 (MAD) to assess the effect of drug on cognitive function.

**MMSE** data will be listed chronologically by cohort/treatment, subject, and visit/day. The classification of MMSE results as normal/abnormal follows the rules in Table 6. Such information will also be included in the listing.

Baseline will be defined as the observation collected at screening. Baseline values, absolute values, and CFB will be summarized by treatment group using standard descriptive statistics. No inferential tests will be conducted on MMSE data.

Table 6. Classification of Normal/Abnormal MMSE Results

| Classification | Description | Rules |
|----------------|-------------------------|-------------------------|
| Normal | No cognitive impairment | Score 24-30 (inclusive) |
| Abnormal | Cognitive impairment | Score <24 |



Study: Study 15-MR-001

# 10 EXPLORATORY ANALYSES

Exploratory assessments will be conducted on blood biomarkers (Th1, Th2 and Th 17 cytokines) in MAD part only. Blood samples will be collected at baseline (Day1, pre-dose), and Day 7 (pre-dose and 4 hrs post dose). See laboratory manual for biomarker processing instructions.

In the descriptive analysis, two types of baselines are considered to calculated CFB values. First, set Day 1 pre-dose value as baseline and calculate CFB for all collection time points after the first dosing on Day 1. Second, set Day 7 pre-dose value as baseline and calculate CFB for the 4-hour post-dose time point on Day 7. Descriptive statistics (number of observations, mean, standard deviation, median, minimum and maximum) will be provided for baseline (Day 1, pre-dose), Day 7 (Pre-dose), change from Baseline to Day 7 (Pre-dose), Day 7 (4 hrs Post-dose), change from Baseline to Day 7 (4 hrs Post-dose) and change from Day 7 (Pre-dose) to Day (4 hrs Post-dose) by treatment.

Paired t-test will be applied on CFB values 1) between Day 1 pre-dose and Day 7 (pre-dose) and 2) between Day 7 pre-dose and Day 7 4 hrs post-dose to determine whether the change within placebo and RP3128 is significant or not.

The CFB values in cytokine expression levels will be compared between placebo and RP3128 using an ANCOVA with the CFB values as the dependent variable, treatment as a fixed effect and corresponding baseline as a covariate. Three different types of CFB will be used: 1) CFB from Day 1 (Pre-dose) to Day 7 (Pre-dose), 2) CFB from Day 1 (Pre-dose) to Day 7 (4 hrs Post-dose), and 3) CFB from Day 7 (Pre-dose) to Day 7 (4 hrs Post-dose). The LSMeans, Standard Errors for each treatment and treatment difference will be presented together with the corresponding 95%-confidence interval and p-value.



Study: Study 15-MR-001

# 11 INTERIM ANALYSES

There is no interim analysis planned in this study. Please note that the results of SAD and MAD will be produced separately. As stated in the protocol, the escalation to next dose level was decided based on the review of blinded safety data from each cohort. Also the dose levels for MAD part was determined based on full blinded safety review of all SAD cohorts. Therefore, the results of the SAD portion of the trial shall have no effect on the MAD), unless there are safety considerations recommended by the Safety Monitoring Committee.


Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### 12 CHANGES TO PLANNED ANALYSES

Due to the nature of the study design of multiple-ascending dose, a few additional endpoints of PK parameters were added to the MAD part.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### 13 APPENDIX:

### APPENDIX A LIST OF CLINICAL LABORATORY TESTS (PART 1-3)

### **Hematology**

• Hemoglobin, Hematocrit, Red blood Cell count, White blood cell count (WBC) with differentials, mean corpuscular volume (MCV), Mean corpuscular hemoglobin (MCH), Mean corpuscular hemoglobin concentration (MCHC), platelet count

### **Coagulation parameters**

• Prothrombin time, Activated partial prothrombin time (APTT)

### **Clinical Chemistry**

- Liver function test: Total bilirubin, Bilirubin (Conjugated and unconjugated), Alkaline Phosphatase, Gamma-GT (GGT), Aspartate aminotransferase (AST), Alanine aminotransferase (ALT),
- Lactate dehydrogenase, Creatinine kinase (CK)
- Kidney function test: Creatinine, Blood Urea nitrogen (BUN), Uric acid
- Lipid profile: Cholesterol, Triglyceride, HDL-Cholesterol, LDL- Cholesterol.
- Total protein, albumin, Glucose
- Electrolytes: Sodium, potassium, calcium, bicarbonates and phosphates

### **Serology (Screening only)**

• HBsAg, Anti-HCV, Anti-HIV 1, 2

### Hormones (Post-menopausal female only) (Screening only)

FSH

### Tuberculin test / QuantiFeron- TB®-Gold test (Screening only)

#### **Pregnancy test (female only)**

- Serum B-HCG
- Urine pregnancy test (UPT) will be performed at later time points in case of suspected pregnancy.

### Alcohol and urine drug screen

- Opiates, methadone, cocaine, amphetamine, cannabinoids, barbiturates and benzodiazepines.
- Alcohol (breath test)

### <u>Urinalysis</u>

• pH, hemoglobin, urobilinogen, ketones, glucose, protein, blood, leukocytes and nitrites



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

## APPENDIX B: PART 1 (SAD) – SCHEDULE OF EVENTS

| | | | | | Assessment pe | eriod | | |
|---|---|---|---|---|---|---|---|---|
| Visits | Screening | | CPU con | finement | | Ambı | ılatory/ follo | w up visit |
| Study Day | -28 to -1 | -1 | 1 | 2 | 3 | 5 | 8 (±1) | 15 (±1) |
| | | Admission | | | (Discharge) | | | $EOS^{14}$ |
| Confinement <sup>1</sup> | | X | X | X | - | - | - | - |
| Ambulatory visits <sup>2</sup> | | - | - | - | - | X | X | X |
| Informed consent <sup>3</sup> | X | | - | - | - | - | - | = |
| Medical history <sup>4</sup> | X | X | - | - | - | X | X | X |
| Demographics <sup>5</sup> | X | - | - | - | - | - | - | - |
| Physical examination <sup>6</sup> | X | X | - | - | X | - | X | X |
| Vital signs <sup>7</sup> | X | X | X | X | X | X | X | X |
| Eligibility assessment | X | X | - | - | - | - | - | - |
| 12-lead ECG <sup>8</sup> | X | X | X | X | X | X | X | X |
| Clinical laboratory <sup>9</sup> | X | X | - | X | X | - | X | X |
| Drug and alcohol screen <sup>10</sup> | X | X | - | - | - | - | - | - |
| HBsAg, HCV, HIV | X | - | - | - | - | - | - | - |
| Tuberculin test / QuantiFeron-<br>TB ®-Gold test | X | | | | | | | |
| Randomization | - | - | X | - | - | = | - | - |
| Pregnancy test (female) 11 | X | X | - | - | - | - | - | - |
| Cognitive test (e.g. MMSE) | X | - | - | - | X | - | - | - |
| Study drug administration | - | - | X | - | - | = | - | - |
| PK sampling blood <sup>12</sup> | - | - | X | X | X | X | X | X |
| Adverse events <sup>13</sup> | X | X | X | X | X | X | X | X |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

| Concomitant medication | X | X | X | X | X | X | X | X |
|------------------------|---|---|---|---|---|---|---|---|

#### Foot notes:

- 1. CPU confinement: subjects will enter the CPU on Day -1 (afternoon) and will be discharged on Day 3 (morning) after safety assessment.
- 2. Ambulatory visit: Day 5, Day 8 and Day 15.
- 3. Informed Consent must be obtained  $\leq$ 28 days prior to the initiation of trial treatment.
- 4. Detailed history will be taken at screening this include present history, past history, allergy, family history, concomitant medication and prior medication (in last 6 weeks); and other medical history. Abbreviated history will be taken at all subsequent visits.
- 5. Demographic will age, sex and race.
- 6. Physical examination includes local and systemic examination and measuring height and weight. Detailed examination will be performed at screening, Day -1, Day 3, Day 8 and Day 15. At other time point, examination will be done as clinically indicated.
- 7. Vitals (temperature, systolic and diastolic blood pressure, respiratory rate and pulse rate) on screening, Day -1 (at the time of admission), Day 1 & Day 2 (pre-dose, 30 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose), Day 3, Day 5, Day 8 and Day 15. At screening, vital signs will be assessed in the supine position after the subject has rested for at least 3 minutes. Blood pressure and pulse will be assessed again after three minutes in the standing position. At other time points, vitals will be measured after 3 minutes supine rest. Vitals should be completed within +/- 30 minute of schedule timing to avoid overlapping; however, in case of adverse events, safety evaluations including vitals and ECGs to be prioritized.
- 8. ECG (single measurement unless stated otherwise): on screening, Day -1 (at the time of admission), Day 1 & Day 2 (pre-dose, 15, 30, 45 min, 1, 2, 4, 6, 8, 12 and 24 hrs post dose), Day 3, Day 5, Day 8 and Day 15. Triplicate ECG will be taken 1 minute apart on screening, Day 1 (pre-dose) and for confirmation of abnormality detected in the single ECG measurement based on Investigator judgement.
- 9. Laboratory assessment: Clinical chemistry, hematology, serum electrolyte, coagulation and urinalysis will be performed. Additionally, FSH will be evaluated at screening to confirm post-menopausal status. Lab investigations will be performed on screening, Day -1, Day 2, Day 3, Day 8 and Day 15. If blood, nitrites or leukocytes are abnormal, automatically microscopic urinalysis will be perform. Additional investigations will be performed if clinically indicated.
- 10. Drug and alcohol screen: This will include screening for opiates, methadone, cocaine, amphetamine, cannabinoids, barbiturates, and benzodiazepines. Alcohol will be screened using alcohol breath test.
- 11. Pregnancy test: β-HCG will be conducted in serum at screening. UPT will be performed at later time points in case of suspected pregnancy.
- 12. PK time points: Day 1 (Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0, 8.0, 12.0, 24.0 and 48 hrs) and at Day 5, Day 8 and Day 15. Window period for sample collection will be outlined in pharmacokinetic manual
- 13. In case of drug related SAE/AE or treatment discontinuation due to adverse event, the subjects will be followed till the resolution/stabilization of the AE or 30 days after the last study dose whichever is the earlier.
- 14. In all subjects, telephone assessments for adverse events and concomitant medications are performed 3 days prior to the EOS visit and as required by physician.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

## APPENDIX C: PART 2 (MAD) — SCHEDULE OF EVENTS

| Study Day | Screen ing | | | | | | | Ass | sessmen | t period | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Adm | ission | CPU Confinement Discha rge | | | | | | | Ambula | tory vis | its | | | |
| Study Day | -60 to -1 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 15 (±1)<br>EOS <sup>18</sup> |
| Confinement <sup>1</sup> | - | X | X | X | X | X | X | X | X | - | - | | - | | | - |
| Ambulatory visits <sup>2</sup> | - | ı | - | - | - | - | - | - | - | - | X | X | X | X | X | X |
| Informed consent <sup>3</sup> | X | | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Medical history <sup>4</sup> | X | X | - | - | - | - | - | - | - | - | X | - | X | - | - | X |
| Demographics <sup>5</sup> | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Physical examination <sup>6</sup> | X | X | - | - | - | X | - | - | - | X | - | - | - | - | - | X |
| Vital signs <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | X | - | X | - | - | X |
| Eligibility assessment | X | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| 12-lead ECG <sup>8</sup> | X | X | X | X | - | - | X | - | X | X | - | - | - | - | - | X |
| Clinical laboratory <sup>9</sup> | X | X | - | X | | - | X | - | X | X | - | - | - | - | - | X |
| Drug and alcohol screen <sup>10</sup> | X | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| HbsAg, HCV, HIV | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Tuberculin test /<br>QuantiFeron- TB<br>®-Gold test | X | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| EEG <sup>11</sup> | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Randomization | - | - | X | - | - | - | - | - | - | - | - | - | - | - | - | - |
| Pregnancy test (female) 12 | X | X | - | - | - | - | - | - | - | - | - | - | _ | - | - | - |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

| Cognitive test (e.g. MMSE) | X | - | - | - | - | - | - | - | - | X | - | - | - | - | - | - |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study drug dispensing <sup>13</sup> | - | - | X | X | X | X | X | X | X | - | - | - | - | - | - | - |
| Study drug administration <sup>14</sup> | - | - | X | X | X | X | X | X | X | - | - | - | - | - | - | - |
| PK sampling blood <sup>15</sup> | - | - | X | X | X | - | X | - | X | X | X | X | X | X | X | X |
| Biomarkers <sup>16</sup> | - | - | X | - | - | - | - | - | X | - | - | - | - | - | - | - |
| Adverse events <sup>17</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

#### Foot notes:

- 1. CPU confinement: Subjects will enter the CPU on Day -1 (afternoon) and will be discharged on day 8 after safety assessment.
- 2. Ambulatory visit: Day 9, Day 10, Day 11, Day 12, Day 13 and Day 15.
- 3. The screening assessments will be performed ≤ 60 days prior to initiation of treatment and informed consent will be obtained prior to initiating any study procedures.
- 4. Detailed history will be taken at screening this include present history, past history, allergy, family history, concomitant medication and prior medication (in last 8 weeks); and other medical history. Abbreviated history will be taken at all subsequent visits.
- 5. Demographic will age, sex and race.
- 6. Physical examination includes local and systemic examination and measuring height and weight. Detailed examination will be performed at screening, Day -1, Day 4, Day 8 and Day 15. At other time point, examination will be done as clinically indicated. Height will only be measured at screening.
- 7. Vitals (temperature, systolic and diastolic blood pressure, respiratory rate and pulse rate) on screening, Day -1 (at the time of admission), Day 1 (pre-dose, 30 min, 1, 2, 4, 6, 12 and 24 hrs post dose), Day 3, Day 4, Day 5, Day 6, Day 7 (pre-dose, 30 min, 1, 2, 4, 6, 12 hrs post dose), Day 8, Day 9, Day 11 and Day 15. At screening, vital signs will be assessed in the supine position after the subject has rested for at least 3 minutes. Blood pressure and pulse will be assessed again after three minutes in the standing position. At other time points, vitals will be measured after 3 minutes supine rest. Vitals should be completed within +/- 30 minute of schedule timing to avoid overlapping; however, in case of adverse events, safety evaluations including vitals and ECGs to be prioritized.
- 8. ECG (single measurement unless stated otherwise): on screening, Day -1 (at the time of admission), Day 1 (pre-dose, 30 min, 1, 2, 4, 6, and 8 hrs post dose), Day 2, Day 5, Day 7 (pre-dose, 30 min, 1, 2, 4, 6, and 8 hrs post dose), Day 8 and Day 15. Triplicate ECG will be taken approximately 1 minute apart on screening and Day 1 (pre-dose). Duplicate repeats will be performed for confirmation of abnormality detected in the single ECG measurement based on Investigator judgement.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

9. Laboratory assessment: Screening, Day -1 (at the time of admission), Day 2 (pre-dose), Day 5 (pre-dose), Day 7 (pre-dose), Day 8 (at discharge) and Day 15. Clinical chemistry, hematology, serum electrolyte, coagulation and urinalysis will be performed. Additionally, FSH will be evaluated at screening to confirm post-menopausal status. If blood, nitrites or leukocytes are abnormal, automatically microscopic urinalysis will be perform. Additional investigations will be performed if clinically indicated.

- 10. Drug and alcohol screen: This will include screening for opiates, methadone, cocaine, amphetamine, cannabinoids, barbiturates, and benzodiazepines. Alcohol will be screened using alcohol breath test.
- 11. EEG will be performed if clinically indicated in case of any symptom.
- 12. Pregnancy test: β-HCG will be conducted in serum at screening. UPT will be performed at later time points in case of suspected pregnancy.
- 13. Study drug (RP3128/placebo) will be dispensed on Day 1 to Day 7.
- 14. Study drug (RP3128/placebo) will be administered once a day from Day 1 to Day 7 at CPU.
- 15. PK time points: Day 1 (Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0, 8.0, 12.0 and 24.0 hr), Day 3, Day 5, Day 7 (Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0, 8.0, 12.0 and 24.0 hrs), Day 9 (48 hrs), Day 10 (72 hrs), Day 11 (96 hrs), Day 12 (120 hrs), Day 13 (144 hrs) and Day 15 (192 hrs). Blood will be collected for PK. Window period for sample collection will be outlined in pharmacokinetic manual.
- 16. Biomarkers: The blood sample will be collected at baseline (Day 1), Day 7 (pre-dose and 4 h post dosing). Measurement of biomarkers (Th1, Th2, and Th17 cytokines) following LPS or CD3/CD28 challenge.
- 17. In case of drug related SAE/AE or treatment discontinuation due to adverse event, the subjects will be followed till the resolution/stabilization of the AE or 30 days after the last study dose whichever is the earlier.
- 18. Window for study assessments: ECG: +/- 15 minutes of the scheduled time; Pre-dose procedures: within 2 hours of dosing.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### 14 TABLE AND LISTING

The following TL shells are provided as a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables and Listings that will be included in the final report. Tables and Listings are numbered following the International Conference on Harmonization (ICH) structure. Table headers, variables names and footnotes will be modified as needed following a review of the blinded data and also following data analyses. Please note that all summary tables and listings will be generated using SAS® Version 9.2 or higher.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.1.1.S/M Disposition of Subjects (SAD/MAD)
Randomized Population

| | Pooled<br>Placebo | RP3128<br>25 mg | RP3128<br>50 mg | RP3128<br>100 mg | RP3128<br>200 mg | RP3128<br>400 mg | Total<br>n (%) |
|---|---|---|---|---|---|---|---|
| Number of Subjects Randomized (N) | XX | XX | XX | XX | XX | XX | XX |
| Number of Subjects in Safety Population (N) | XX | XX | XX | xx | xx | XX | XX |
| Number of Subjects in PK Population [n (%)] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects who Completed the Study [n (%)] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects who Discontinued Early [n (%)] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Allergic Reaction / Anaphylaxis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Concomitant Medication Interfering W/ PK | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Emesis Within 10 hrs Post Dose | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to Follow-up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Physician Decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Study Terminated by Sponsor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal by Subject | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are calculated based on the number of subjects in the Safety population per treatment group and overall.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.1.2.S/M Summary of Demographics (SAD/MAD) Safety Population

| | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>50 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) | RP3128<br>400 mg<br>(N=xx) | All Subjects (N=xx) |
|---|---|---|---|---|---|---|---|
| Age (years)* | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx | XX.XX |
| Minimum | XX | xx | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | xx | XX | XX | XX | XX | XX |
| Sex, n (%) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>\*</sup>Age at Informed Consent

Note: Percentages are calculated based on the number of subjects in the Safety population per treatment group and overall.

Programming Note: Table will also include race, ethnicity, height (cm), weight (kg), and BMI (kg/m2).



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.1.3.M Summary of Drug Administration (MAD) Safety Population

| | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>400 mg<br>(N=xx) |
|---|---|---|---|---|
| Number (%) of subjects who received all doses | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number of Days on Treatment | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.2.1.1.X.S RP3128 Plasma Concentrations (ng/mL) by Time Point (SAD) Safety Population <Dose Level>

| | | | | | | | | Time | Point | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cohort<br>/Subject | 0h | 0.25h | 0.5h | 1h | 2h | 4h | 6h | 8h | 12h | 24h | 48h | 96h | 168h | 336h |
| | XXXX | XXX.X | XXX,X | XXX,X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | xxx.x | XXX.X |
| Statistics | | | | | | | | | | | | | | | |
| N | | XX | XX | XX | xx | XX | XX | XX | XX | xx | XX | XX | XX | XX | xx |
| Mean <sup>1</sup> | | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx |
| CV (%) | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | | xxx | xxx | xxx | Xxx | Xxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx |
| Median | | xxx.x | xxx.x | xxx.x | xxx.x | XXX.X | XXX.X | xxx.x | xxx.x | xxx.x | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x |
| Maximum | | XXX | XXX | XXX | Xxx | Xxx | XXX | XXX | XXX | XXX | xxx | xxx | xxx | xxx | xxx |

N= Number of subject for which plasma sample was collected at each time point.

Programming Note: X will be assigned as 1, 2, 3.... as per each RP3128 dose level. Time point may vary depending on the actual number of sample collection.

<sup>&</sup>lt;sup>1</sup>Mean calculated based on number of subjects (N).

<sup>&</sup>lt;Dose Level> = RP3128 25 mg, 50 mg, 100 mg, 200 mg, 400 mg in SAD



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Table 14.2.1.1.1.X.M RP3128 Plasma Concentrations (ng/mL) by Time Point (MAD) – Day 1 Safety Population <Dose Level>

| | | | | | | Time | Point | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cohort<br>/Subject | 0h | 0.25h | 0.5h | 1h | 2h | 4h | 6h | 8h | 12h | 24h |
| | XXXX | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Statistics | | | | | | | | | | | |
| N | | xx | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| Mean <sup>1</sup> | | XXX.X | xxx.x | XXX.X | XXX.X | xxx.x | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |
| SD | | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV (%) | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | | xxx | XXX | xxx | Xxx | Xxx | XXX | XXX | XXX | XXX | XXX |
| Median | | XXX.X | xxx.x | XXX.X | XXX.X | xxx.x | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |
| Maximum | | xxx | XXX | XXX | Xxx | Xxx | XXX | XXX | xxx | XXX | XXX |

N= Number of subject for which plasma sample was collected at each time point.

Programming Note: X will be assigned as 1, 2, 3.... as per each RP3128 dose level. Time point may vary depending the actual data.

<Dose Level> = RP3128 25mg, 100mg, 400mg in MAD

<sup>&</sup>lt;sup>1</sup>Mean calculated based on number of subjects (N).



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.2.1.1.2.X.M RP3128 Plasma Concentrations (ng/mL) by Time Point (MAD) – Day 7 Safety Population <Dose Level>

| | | Time Point | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cohort /Subject | 0h | 0.25h | 0.5h | 1h | 2h | 4h | 6h | 8h | 12h | 24h | 48h | 72h | 96h | 120h | 144h | 192h |
| | XXXX | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | xxx.x | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | xxx.x | XXX.X | xxx.x | xxx.x |
| Statistics | | | | | | | | | | | | | | | | | |
| N | | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean <sup>1</sup> | | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| CV (%) | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | | XXX | XXX | XXX | Xxx | Xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Median | | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X |
| Maximum | | XXX | XXX | XXX | Xxx | Xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

N= Number of subject for which plasma sample was collected at each time point.

Programming Note: X will be assigned as 1, 2, 3.... as per each RP3128 dose level. Time point may vary depending the actual data.

<Dose Level> = RP3128 25mg, 100mg, 400mg in MAD

<sup>&</sup>lt;sup>1</sup>Mean calculated based on number of subjects (N).



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.2.1.2.X.S RP3128 – Summary of PK Parameters (SAD)
PK Population
<Dose Level>

| Cohort/Subject | $AUC_{0-t}$ | $AUC_{0-inf}$ | $C_{max}$ | $T_{max}$ | $K_{el}$ | $T_{1/2}$ |
|---|---|---|---|---|---|---|
| · | (h*ng/mL) | (h*ng/mL) | (ng/mL) | (h) | (1/h) | (h) |
| XXXX | XXX | Xxx | XXX | XXX | XXX | XXX |
| xxxx | XXX | Xxx | XXX | XXX | XXX | XXX |
| | XXX | Xxx | XXX | XXX | XXX | XXX |
| Statistics | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XXX | XXX | XXX | XXX | XXX | XXX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Maximum | XXX | XXX | XXX | XXX | XXX | XXX |
| Geo Mean <sup>1</sup> | XXX.X | XXX.X | XXX.X | NA | NA | NA |
| Geometric CV% | XX.X | XX.X | XX.X | NA | NA | NA |

N=Number of subjects with derivable PK parameter.

Programming Notes: Geometric mean shall be calculated for all PK parameters except  $T_{max}$ ,  $t_{1/2}$  and  $K_{el}$ .  $T_{max}$  will only have n, median, min, max provided.

X will be assigned as 1, 2, 3.... as per each RP3128 dose level.

<sup>&</sup>lt;Dose Level> = RP3128 25 mg, 50 mg, 100 mg, 200 mg, 400 mg



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.2.1.2.1.X.M RP3128 – Summary of PK parameters (MAD) – Day 1
PK Population
<Dose Level>

| Cohort/Subject | C <sub>max</sub> | AUC <sub>0-24</sub><br>(ng·h/mL) | T <sub>max</sub> | T <sub>1/2</sub> |
|---|---|---|---|---|
| | (ng/mL) | (lig'ii/liiL) | (h) | (h) |
| XXXX | XXX | XXX | XXX | XXX |
| XXXX | XXX | XXX | XXX | XXX |
| Statistics | | | | |
| N | XX | XX | XX | XX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| CV (%) | XX.X | XX.X | XX.X | XX.X |
| Minimum | XXX | X.X | X.X | X.X |
| Median | XXX.X | XX.X | XX.X | XX.X |
| Maximum | XXX | X.X | X.X | X.X |
| Geo Mean <sup>1</sup> | XXX.X | XXX.X | NA | NA |
| Geometric CV% | XX.X | XX.X | NA | NA |

N=Number of subjects with derivable PK parameter.

Programming Note: <Dose Level> = RP3128 25mg, 100mg, and 400mg.

X will be assigned as 1, 2, and 3 as per each RP3128 dose level.

<sup>&</sup>lt;sup>1</sup>: Geo Mean: Geometric means are based on the arithmetic means of ln-transformed values



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Table 14.2.1.2.2.X.M RP3128 – Summary of C<sub>trough</sub> (MAD) PK Population <Dose Level>

| Caland Caland | | $C_{trough}$ (ng/mL) | |
|-----------------------|--------|----------------------|--------|
| Cohort/Subject | Day 3 | Day 5 | Day 7 |
| XXXX | XXX | XXX | XXX |
| xxxx | xxx | XXX | XXX |
| Statistics | | | |
| N | XX | XX | xx |
| Mean | XXX.X | XXX.X | xxx.x |
| SD | XXX.XX | XXX.XX | XXX.XX |
| CV (%) | XX.X | XX.X | XX.X |
| Minimum | XXX | XXX | X.X |
| Median | XXX.X | XXX.X | XX.X |
| Maximum | XXX | XXX | X.X |
| Geo Mean <sup>1</sup> | XXX.X | XXX.X | xxx.x |
| Geometric CV% | XX.X | XX.X | xx.x |

N=Number of subjects with derivable PK parameter.

Programming Note: <Dose Level> = RP3128 25mg, 100mg, and 400mg.

X will be assigned as 1, 2, and 3 as per each RP3128 dose level.

<sup>&</sup>lt;sup>1</sup>: Geo Mean: Geometric means are based on the arithmetic means of ln-transformed values



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.2.1.2.3.X.M RP3128 – Summary of PK parameters (MAD) – Day 7
PK Population
<Dose Level>

| Cohort/Subject | $C_{max}$ (ng/mL) | C <sub>min</sub> (ng/mL) | AUC <sub>0-24</sub><br>(ng·h/mL) | Cav<br>(ng/mL) | Degree of Fluctuation | Swing | T <sub>max</sub> (h) | T <sub>1/2</sub> (h) |
|---|---|---|---|---|---|---|---|---|
| XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Statistics | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum | XXX | XXX | X.X | XXX | XXX | X.X | X.X | X.X |
| Median | XXX.X | XXX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XXX | XXX | X.X | X.X | X.X | X.X | X.X | X.X |
| Geo Mean <sup>1</sup> | XXX.X | XXX.X | XXX.X | XXX.X | NA | NA | NA | NA |
| Geometric CV% | XX.X | XX.X | XX.X | XX.X | NA | NA | NA | NA |

N=Number of subjects with derivable PK parameter.

Programming Note: <Dose Level> = RP3128 25mg, 100mg, and 400mg

X will be assigned as 1, 2, and 3 as per each RP3128 dose level.

<sup>1:</sup> Geo Mean: Geometric means are based on the arithmetic means of ln-transformed values



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.2.2.X.1.M Summary of Cytokines <expression value>: Change from Baseline (MAD)

Safety Population

| | | Safety Popu | |
|---|---|---|---|
| | | Placebo | eatment RP3128 |
| Visit and Time Point | Statistic | (N=xx) | (N=xx) |
| Baseline (Day 1, Pre-dose) | | *** | *** |
| | n<br>Mean ± SD | $Xx \\ xx.x \pm x.xx$ | $Xx \\ xx.x \pm x.xx$ |
| | Median | XX.X = X.XX $XX.X$ | XX.X |
| | Min, Max | XX , XX | XX , XX |
| Day 7 (Pre-dose) | | | |
| | n<br>Mean ± SD | $\begin{array}{c} xx \\ xx.x \pm x.xx \end{array}$ | $Xx \\ xx.x \pm x.xx$ |
| | Median | $XX.X \perp X.XX$ $XX.X$ | $XX.X \perp X.XX$<br>XX.X |
| | Min, Max | XX, XX | XX , XX |
| Change from Baseline <sup>1</sup> | | | |
| _ | n<br>Maan SD | XX | Xx |
| | Mean ± SD<br>Median | $xx.x \pm x.xx$<br>xx.x | $XX.X \pm X.XX$<br>XX.X |
| | Min, Max | XX, XX | XX , XX |
| | Paired t-test | X.XX | x.xx |
| Day 7 (4 hr Post-dose) | | | |
| Change from Baseline <sup>1</sup> | | | |
| Change from Baseline <sup>2</sup> | | | |

Note: 1 Baseline set at Day 1 pre-dose; 2 baseline set at Day 7 pre-dose

Data source: Listings 16.2.6.1

Programming note: Replace <expression value> with Th1, Th2, and Th17 and X will be assigned as 1, 2, and 3 for expression Th1, Th2 and Th17 respectively



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.2.2.X.2.M ANCOVA Results of Cytokine <expression value> Change from Baseline to Day 7 (Pre-dose/Post-dose)/ Difference between Pre-dose and Post-dose on Day 7 (MAD)

Safety Population

| | | | | | | Difference b | etween RP3128 to Pla | icebo | |
|---|---|---|---|---|---|---|---|---|---|
| Item | Treatment | n | LSMeans Std Err | | LSMeans | Std Err | 95%-confidence<br>Interval | P-value<br>Treatment | P-value<br>Baseline |
| CFB Day 7 (Pre-dose) | Overall | XXX | | | | | | X.XXXX | X.XXXX |
| | Placebo | XXX | x.xxx | X.XXX | | | | | |
| | RP3128 | XXX | x.xxx | X.XXX | X.XXX | X.XXX | x.xxx, x.xxx | X.XXXX | |
| CFB <sup>1</sup> Dav 7 (4 hr Post-dose) | Overall | XXX | | | | | | X.XXXX | x.xxxx |
| | Placebo | xxx | X.XXX | x.xxx | | | | | |
| | RP3128 | XXX | x.xxx | X.XXX | X.XXX | x.xxx | x.xxx, x.xxx | X.XXXX | |
| CFB <sup>2</sup> Day 7(4 hr Post dose) | | | | | | | | | |

Note: 1 Baseline set at Day 1 pre-dose 2 Baseline set at Day 7 pre-dose

LSMeans: Least square means; Std Err: Standard error

LSMeans, Std Err, 95% confidence intervals and p-values are based on an ANCOVA with change from baseline as dependent variable, visit and treatment as fixed effect and baseline as covariate. P-values are from two-sided test at 5%-level.

Data source: Listings 16.2.6.1

Programming note: Replace <expression value> with Th1, Th2, and Th17 and X will be assigned as 1, 2, and 3 for expression Th1, Th2 and Th17 respectively



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.3.1.1.S/M Treatment-Emergent Adverse Events – Overall Summary (SAD/MAD) Safety Population

| | | | Treatmen | at at Onset of Adver | se Event | | _ |
|---|---|---|---|---|---|---|---|
| | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>50 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) | RP3128<br>400 mg<br>(N=xx) | RP3128<br>Overall<br>(N=xx) |
| Number (%) of Subjects with TEAE | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Number (%) of Subjects with Serious TEAE | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Number (%) of Subjects with Severe TEAE | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Number (%) of Subjects with Related TEAE | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Number (%) of Subjects with Study Discontinued due to TEAE | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |

Notes: A treatment-emergent adverse event (TEAE) is an AE, which starts or worsens after treatment with the study drug.

An AE is considered to be related if it is reasonably related to study treatment.

Summaries are presented as: number of subjects (percentage of subjects) [number of events]



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.3.1.2.S/M Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (SAD/MAD)
Safety Population

| | | Treatmen | nt at Onset of Advers | e Event | | | |
|---|---|---|---|---|---|---|---|
| System Organ Class/<br>Preferred Term | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>50 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) | RP3128<br>400 mg<br>(N=xx) | RP3128<br>Overall<br>(N=xx) |
| Any System Organ Class | | | | | | | |
| Any Event | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Cardiac Disorders | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Any Event | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Bradycardia | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |

...

Notes: A treatment-emergent adverse event (TEAE) is an AE, which starts or worsens after treatment with the study drug.

For each row category, a subject with two or more adverse events in that category is counted only once.

Summaries are presented as: number of subjects (percentage of subjects) [number of events]



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.3.1.3.S/M Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Intensity (SAD/MAD) **Safety Population** 

| | | | Treatment at On | set of Adverse Eve | ent | | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class/<br>Preferred Term | Maximum<br>Intensity | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>50 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) | RP3128<br>400 mg<br>(N=xx) | RP3128<br>Overall<br>(N=xx) |
| Any System Organ<br>Class | | | | | | | | |
| Any Event | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Cardiac Disorders | | | | | | | | |
| Any Event | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: A treatment-emergent adverse event (TEAE) is an AE which starts or worsens after treatment with the study drug.

For each row category, a subject with two or more adverse events in that category is counted only once at the maximum severity level.

Summaries are presented as: number of subjects (percentage of subjects)



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.3.1.4.S/M Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Relationship (SAD/MAD)
Safety Population

| | | Treatment a | t Onset of Adv | erse Event | | | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class/<br>Preferred Term | Maximum Relationship | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>50 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) | RP3128<br>400 mg<br>(N=xx) | RP3128<br>Overall<br>(N=xx) |
| Any System Organ<br>Class | | | | | | | | |
| Any Event | No Reasonable Possibility | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Reasonable Possibility | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Cardiac Disorders | | | | | | | | |
| Any Event | No Reasonable Possibility | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Reasonable Possibility | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: A treatment-emergent adverse event (TEAE) is an AE which starts or worsens after treatment with the study drug.

For each row category, a subject with two or more adverse events in that category is counted only once at the maximum relationship level. Summaries are presented as: number of subjects (percentage of subjects)



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.3.3.1.X.S/M Summary of <laboratory Panel> (SAD/MAD) Safety Population

### Example of quantitative data:

| Parameter<br>(unit) | Statistic | Pooled<br>Placebo | RP3128<br>25 mg | RP3128<br>50 mg | RP3128<br>100 mg | RP3128<br>200 mg | RP3128<br>400 mg |
|---|---|---|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Albumin (g/L) Baseline* | | | | | | | |
| , | Summary Statistics | | | | | | |
| | n | XX | XX | XX | XX | XX | Xx |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | XX | Xx |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | Relation to Reference Range, n (%) | | | | | | |
| | n | n | n | n | n | n | n |
| | Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | Low | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | High | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Day X | | | | | | | |
| CFB on Da | y X | ••• | | | | | |

Note: CFB = Change from Baseline

\*Baseline is defined as the last observation prior to dosing on Day 1.

<Laboratory Panel> = Hematology, Chemistry, Urinalysis

Programming Note: X will be assigned as 1, 2, and 3 as per laboratory panels. Day X will depends on SAD or MAD;

Relation to Reference Range will be summarized for raw data only, not for change-from-baseline values



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Example of qualitative data:

| Parameter (unit) | Visit | | Pooled | RP3128 | RP3128 | RP3128 | RP3128 | RP3128 |
|---|---|---|---|---|---|---|---|---|
| | | | Placebo | 25 mg | 50 mg | 100 mg | 200 mg | 400 mg |
| | | | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Urine Protein (G/L) | Baseline* | | | | | | | |
| | | Frequency, n (%) | | | | | | |
| | | n | n | n | n | n | n | n |
| | | Category 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Category 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Relation to Reference Range, n (%) | | | | | | |
| | | n | n | n | n | n | n | n |
| | | Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Day X | | ••• | | | | | |
| | Follow-up or<br>ET | | | | | | | |
| •••• | | | | | | | | |

<sup>\*</sup>Baseline is defined as the last observation prior to dosing on Day 1.

Notes: Percentages are calculated based on the number of subjects in the Safety population per treatment group.

Programming Note: X will be assigned as 1, 2, 3 as per laboratory panels.

<sup>&</sup>lt;Laboratory Panel> = Hematology, Chemistry, Urinalysis



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.3.3.2.X.S/M <Laboratory Panel>: Shift Table from Baseline to End of Treatment Results (SAD/MAD)

Safety Population

| | | | Baseline (n=xx)* | | | |
|---|---|---|---|---|---|---|
| Laboratory Parameter (unit) | Study Day<br>[Treatment] | Parameter | Low | Normal | High/Abnormal# | Total |
| Parameter 1 (unit) | Day 3/8 [Placebo] | Low | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | High | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Day 3/8 [RP3128 25 mg] | •••• | ••• | | | |
| | | •••• | | | | |
| •••• | | | | | | |

Note: Doses are Total Daily Dose.

Notes: \*Baseline is defined as the last observation prior to dosing on Day 1.

# For categorical assays, abnormal results are counted under the "High/Abnormal" column ('Low' column is 'N/A')

Note: Percentages are calculated based on the number of subjects in the Safety population per treatment group.

Note: <Laboratory Panel> = Hematology, Chemistry, Urinalysis

Programming Note: Table will continue for other lab parameters. X will be assigned as 1, 2, 3 as per laboratory panels. For SAD, Day 3 will be used to compare with Baseline. For MAD, Day 8 will be used.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.3.4.X.S/M Summary of Vital Signs Data by Treatment, Visit and Time Point (SAD/MAD) Safety Population

<Vital Signs Parameter (unit)>

| Time Point/<br>Visit (Day) | Statistic | Pooled<br>Placebo | RP3128<br>25 mg | RP3128<br>50 mg | RP3128<br>100 mg | RP3128<br>200 mg | RP3128<br>400 mg |
|---|---|---|---|---|---|---|---|
| D 1: * | | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline* | | | | | | | |
| | n | XX | XX | XX | XX | XX | Xx |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | XX | Xx |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX | Xx |

0.5h Day 1 0.5h Day 1 CFB

. . .

Note: CFB = Change from Baseline

Programming Note: Table also includes all days and time points except screening and check-in.

X will be assigned as 1, 2, 3, 4 and 5 as per vital sign parameters (unit).

<sup>\*</sup>Baseline is defined as the last observation prior to the dose on Day 1.

<sup>&</sup>lt;Vital Signs Parameter (unit)> = Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg), Heart Rate (bpm), Respiratory Rate (breaths/min), Oral Temperature (°C)



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.3.4.6.S/M Summary of Weight Data by Treatment and Time Point (SAD/MAD) Safety Population

| Time Point | Statistic | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>50 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) | RP3128<br>400 mg<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Check-in | | | | | | | |
| (Baseline) | | | | | | | |
| | n | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX | XX |

Day 3/4

Day 3/4 CFB

Day 8

Day 8 CFB

Day 15

Day 15 CFB

Note: CFB = Change from Baseline

Programming Note: For SAD, Day 3 will be applied. For MAD, Day 4 will be applied.

<sup>\*</sup>Baseline is defined as the last observation prior to the dose on Check-in.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Table 14.3.5.1.S/M Summary of Overall ECG Interpretation (SAD/MAD) Safety Population

| | | surety 1 opu | | | | |
|---|---|---|---|---|---|---|
| | Pooled<br>Placebo<br>(N=xx) | RP3128<br>25 mg<br>(N=xx) | RP3128<br>50 mg<br>(N=xx) | RP3128<br>100 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) | RP3128<br>200 mg<br>(N=xx) |
| Baseline | | | | | | |
| n | XX | XX | XX | xx | XX | Xx |
| Normal, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, Not Clinically Significant, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, Clinically Significant, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Follow-up or ET | | | | | | |
| n | XX | XX | XX | XX | XX | Xx |
| Normal, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, Not Clinically Significant, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, Clinically Significant, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing, n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are calculated based on the number of subjects in the Safety population per treatment group.

Programming Note: Table also includes time points and visits listed in the section 9.5



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.3.5.X.S/M Summary of ECG Continuous Data (SAD/MAD) Safety Population

<ECG Parameter (unit)>

| | | \ECG i ai a | iniciei (unit) | | |
|---|---|---|---|---|---|
| Time Point/<br>Statistic | Pooled<br>Placebo<br>(N=xx) | RP3128<br>20 mg<br>(N=xx) | RP3128<br>60 mg<br>(N=xx) | RP3128<br>120 mg<br>(N=xx) | RP3128<br>240 mg<br>(N=xx) |
| Baseline* | | | | | |
| n | XX | XX | XX | XX | Xx |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | Xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | Xx |
| 5 min | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| ••• | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX |
| 5 min CFB | | | | | |

CFB = Change from Baseline

Note: \*Baseline is defined as the last observation prior to the dose.

<ECG Parameter (unit)> = Ventricular Rate (bpm), PR interval (msec), QRS duration (msec), QT Interval (msec), QTcB Interval (msec)

Programming Note: Table also includes time points and visits listed in the section 9.5

X will be 2, 3, 4, 5 and 6 for VR, PR, QRS, QT and QTcB.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Table 14.3.6.1.S/M Summary of Mini-Mental State Examination (SAD/MAD) Safety Population

| Visit/Statistic | Pooled | RP3128 | RP3128 | RP3128 | RP3128 | RP3128 |
|-----------------|---------|--------|--------|--------|--------|--------|
| | Placebo | 25 mg | 50 mg | 100 mg | 200 mg | 400 mg |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline* | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX |
| Day 3/8 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX |
| Day 3/8 CFB | | | | | | |
| ••• | | | | | | |

CFB = Change from Baseline

Note: \*Baseline is defined as the observation from screening.

Programming Note: Day 3 will be used for SAD and Day 8 will be used for MAD.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Listing 16.1.7.S/M Randomization Scheme and Code (SAD/MAD) Randomized Population

| Randomization<br>Number | Cohort/Treatment | Age*<br>(years) | Date of Randomization | Sex |
|---|---|---|---|---|
| xxxx | 1/Placebo | 30 | DDMONYYYY | F |

<sup>\*</sup>Age at Informed Consent



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.1.S/M Subject Disposition and Completion/Discontinuation (SAD/MAD) **Randomized Population**

| Cohort/<br>Treatment | Subject | Completed<br>Study | Date of Study Completion<br>or Early Discontinuation /<br>Date of last Contact | Date of dosing | Reason for Study<br>Discontinuation* |
|---|---|---|---|---|---|
| 1/Placebo | xxxx | Yes | DDMONYYYY/<br>DDMONYYYY | DDMONYYYY | xxxxxxxxxx |

<sup>\*</sup>A corresponding AE number will be displayed if Reason for Treatment Discontinuation or Reason for Study Discontinuation is "Adverse Event".



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.2.S/M Protocol Deviations (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Start Date of deviation | Visit/Day | Description of Protocol Deviation | Classification | Category |
|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | DDMONYYYY | xxxx | Xxxxxx | Major/Minor | Procedures/Assessments<br>Outside Protocol Window |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Listing 16.2.3.S/M Exclusions from Analysis Populations (SAD/MAD) Randomized Population

| Cohort/<br>Treatment | Subject | Excluded from Safety Population | Reason for Exclusion from the Safety Population | Excluded from PK Population | Reason for Exclusion from the PK Population |
|---|---|---|---|---|---|
| 1/Placebo | xxxx | No | Xxxxxxx | Yes | Xxxxxxx |
| ••• | | | | | |


Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.4.S/M Demographics and Informed Consent at Screening (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Informed<br>Consent Date | Sex | Date of Birth | Age*<br>(years) | Race | Ethnicity | Height (cm) | Weight (kg) | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|---|---|
| 1/Placebo | XXXX | DDMONYYYY | X | DDMONYYYY | XX | XXXXX | xxxxx | XXX | XX | XX |

...

<sup>\*</sup>Age at Informed Consent



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.5.1.S/M Study Drug Administration and Compliance (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Visit/Day | Study Drug<br>Administered? | Route of Administration | Dose/Unit | Start date | Start time/End time | Treatment<br>Comment |
|---|---|---|---|---|---|---|---|---|
| 1/Placebo | XXXX | Day 1 | Yes | Oral | xx/mg | DDMONYYYY | HH:MM/HH:MM | XXXXXXXX |

. . .



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.5.2.S/M Pharmacokinetic Sample Collection Data (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Dosing Date and<br>Time | Date of Sample<br>Collection | Scheduled<br>Time Point (hr) | Elapsed Time*<br>(hr)* | Actual Sample<br>Collection Time<br>(HH:MM) | Time<br>Deviation**<br>(min) | Plasma<br>Concentration<br>(ng/mL) |
|---|---|---|---|---|---|---|---|---|
| 1/RP3128<br>20 mg | xxxx | DDMONYYYY<br>HH:MM | DDMONYYYY | Pre-dose | -1.4 | HH:MM | xx | XX |
| | | | | 0.083 | 0.083 | HH:MM | XX | XX |
| | | | | 0.25 | 0.25 | HH:MM | XX | XX |
| | | | | 0.5 | 0.51 | HH:MM | XX | XX |
| | | | | 2 | 2.1 | HH:MM | XX | XX |
| | | | | 6 | 6 | HH:MM | XX | XX |
| | | | | 12 | 12 | HH:MM | XX | XX |

<sup>\*</sup>Difference between actual sample collection time and dosing time

Note: BLQ = Below the limit of quantification.

Note: HH:MM = Hours: Minutes

<sup>\*\*</sup>Difference actual collection and scheduled collection time (post treatment time points only)



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.5.3.S Pharmacokinetic Parameters (SAD) PK Population

| Cohort/Treatment | Subject | Lower<br>Time*<br>(h) | Upper<br>Time*<br>(h) | Number of points used in $K_{el}$ estimation | Adjusted<br>R-Square | K <sub>el</sub> (1/h) | t <sub>1/2</sub> (h) |
|---|---|---|---|---|---|---|---|
| 1/RP3128 25 mg | xxxx | xxx | xxx | xxx | xxx | xxx | xxx |

<sup>\*</sup>Lower time and upper time are the lower and upper limits on time, respectively, for values to be included in the estimation of Kel. Note: Minimum 3 points will be used to estimate Kel.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.5.4.S/M Reasons Why Pharmacokinetic Parameters Could Not be Determined (SAD/MAD)

| Cohort/Treatment | Subject | Pharmacokinetic Parameter (Units) | Original<br>Value | Reason |
|---|---|---|---|---|
| 1/RP3128 20 mg | xxxx<br> | K <sub>el</sub> (h) | xxx | Xxxxxxxxx |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.6.1: Cytokine assessment

| | | | | | | Cytokine | Test |
|---|---|---|---|---|---|---|---|
| Cohort/Treatment | Subject | Time<br>Visit Date Point | | <br>Th1 | Th2 | Th17 | |
| 1/Placebo | 1001 | Day 1 | DDMMMY | YYY Pre-dose | XX | XX | XX |
| | | Day 7 | DDMMMY | YYYY Pre-dose | XX | XX | XX |
| | | Day 7 | DDMMMY | YYYY post-dose | XX | XX | XX |
| 2/RP3128 25mg | xxxx | | | | | | |

Programming Note: the list of cytokine here is just an example, the final listing will show all cytokines available in the eCRF.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.7.1.S/M Adverse Events (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Visit | <b>A</b><br>E<br># | System Organ<br>Class/<br>Preferred<br>Term/<br>Verbatim Term | TE<br>AE<br>? | Ongo<br>-ing? | Start Date and<br>Time/<br>Stop Date and<br>Time/ | Time from<br>Dosing/<br>Duration<br>(DD:HH:MM)* | Toxicity<br>Grade ( if<br>applicable) | Severity/<br>Serious/<br>Relationship to<br>Study Drug/<br>Outcome | Study Drug<br>Action Taken/<br>Non-Drug<br>Action Taken | Caused<br>Study<br>Disconti<br>nuation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | х | Gastrointestina<br>l disorders/<br>Vomiting/<br>Vomiting | Y | Y | DDMONYYYY<br>HH:MM | DD:HH:MM/<br>DD:HH:MM | 2 | Moderate/ No/<br>Related /<br>Recovered/Res<br>olved | Not Applicable/<br>None | |

\*DD:HH:MM = Days:Hours:Minutes



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.7.2.S/M Deaths, Other Serious and Significant Adverse Events Safety Population (SAD/MAD)

| Cohort/<br>Treatment | Subject | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Date and Time of Event/<br>Date and Time of<br>Resolution | Severity/ Serious/<br>Relationship to Study Drug/<br>Outcome | Study Drug Action<br>Taken/ Other Action<br>Taken |
|---|---|---|---|---|---|
| 1/Placebo | xxxx<br> | Nervous system disorders/<br>Migraine/ Migraine | DDMONYYYY HH:MM/<br>DDMONYYYY HH:MM | Mild/ No/ Possibly Related/<br>Recovered/Resolved | Dose Not Changed/<br>ConMed Taken (CM #<br>1) |

Programming Note: this listing will only be produced when any SAE has occurred during the study.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.8.X.S/M < Laboratory Panel> (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Visit/Day | Date of Sample<br>Collection | Lab test (Unit) | Value | Reference<br>Range<br>Indicator | Normal<br>Range | Completion<br>Status |
|---|---|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | Screening | DDMONYYYY | Xxxxxxxxxxxxxxxxx(xxxx) | XX | High | xx - xxx | Yes |
| | | | | Xxxxxxxxxxxxxxxxx(xxxx) | XX | Abnormal | Negative | Yes |
| | ••• | | | | | | | |

<Laboratory Panel> = Hematology, Chemistry, Urinalysis

Note to programmer: X will be assigned as 1, 2, and 3 as per each laboratory panels.

### Listing 16.2.8.X.S/M <Laboratory Panel>: Abnormal Results (SAD/MAD) Safety Population

| Cohort/Treatment Subject Visit/Day Date/Time Lab test (Unit) Value Reference Normal Significance# | Cohort/Treatment | Subject | Visit/Day | Date/Time | Lab test (Unit) | Value | Reference | Normal | Significance# |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

| | | | | | | Range<br>Indicator | Range | |
|---|---|---|---|---|---|---|---|---|
| 1/Placebo | XXXX | Screening | DDMONYY<br>YY HH:MM | xxxxxxx | X.X | Abnormal | Negative | NCS |
| | | | | | | High | xx-xxx | CS |

Note: #Significance: CS = Clinically Significant, NCS = Not Clinically Significant

<Laboratory Panel> = Hematology, Chemistry, Urinalysis
Note to programmer: X will be assigned as 4, 5, and 6 as per each laboratory panels.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.8.7.S/M Viral Screen and TB Test at Screening (SAD/MAD) Safety Population

| Cohort/Treatment | Subject | Date and Time | Hepatitis B Surface<br>Antigen | Hepatitis C Virus<br>Antibody | HIV 1/2 Antibody | Tuberculin test<br>/QuantiFeron-TB - Gold test |
|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | DDMONYYYY<br>HH:MM | Negative | Negative | Non-Reactive | Negative |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.8.8.S/M Drug and Alcohol Screen (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Visit | Collection<br>Date | Opiates | Methadone | Cocaine | Amphe tamine | Cannabinoids | Barbiturate | Benzodia<br>-zepine | Alcohol Breath<br>Test |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | Screening | DDMON<br>YYYY | Negative | Negative | Positive | Negative | Negative | Negative | Negative | Negative |
| | | Day -1 | | | | | | | | | |
| | •••• | | | | | | | | | | |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.9.1.S/M Vital Signs (SAD/MAD) Safety Population

| Cohort/Treat ment | Subject | Visit | Time<br>Point | Position | Date | Time | SBP<br>(mmH<br>g) | DBP<br>(mmH<br>g) | HR<br>(bpm) | RR<br>(bpm) | Temp<br>(°C) | Weight (kg) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | Screening | | Supine | DDMONY<br>YYY | HH:M<br>M | XXX | XX | XX | XX | XX | xx |
| | | Check-in<br>Day -1 | | | DDMONY<br>YYY | HH:M<br>M | XXX | XX | XX | XX | XX | XX |
| | | Day 1 | Pre-dose | | DDMONY<br>YYY | HH:M<br>M | XXX | XX | XX | XX | XX | |
| | | | 30 min | | DDMONY<br>YYY | HH:M<br>M | XXX | XX | XX | XX | XX | |
| | | | 1 hour | | DDMONY<br>YYY | HH:M<br>M | XXX | XX | XX | XX | XX | |
| | | Day 2 | | | | | | | | | | |
| | | Follow-<br>up or ET | | | | | | | | | | |

.....

Note: SBP = Systolic Blood Pressure; DBP = Diastolic Blood Pressure; HR = Heart Rate; RR = Respiration Rate; Temp = Oral Temperature; bpm = Beats per Minute or Breaths per Minute



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.10.1.S/M Electrocardiogram (ECG) (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Visit | Time<br>Point | Date and<br>Time | Was the ECG Performed ? | ECG Overall<br>Interpre-<br>tation | VR<br>(bpm) | PR (msec) | QRS<br>(msec) | QT (msec) | QTcB<br>(msec) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | Screening | | DDMONYYYY<br>HH:MM | Yes | Abnormal/NCS | XX | xxx | XX | XX | XXX |
| | | Day 1 | Pre-dose | DDMONYYYY<br>HH:MM | No | | | | | | |
| | | | 15 min | DDMONYYYY<br>HH:MM | Yes | Normal | XX | XXX | XX | XX | xxx |
| | | | 30 min | DDMONYYYY<br>HH:MM | NU | | | | | | |
| | | | 45 min | DDMONYYYY<br>HH:MM | Yes | Normal | XX | XXX | XX | XX | xxx |
| | | | 1 hour | DDMONYYYY<br>HH:MM | Yes | Normal | XX | XXX | XX | XX | XXX |
| | | Day 3 | | DDMONYYYY<br>HH:MM | Yes | Normal | xx | xxx | xx | xx | XXX |
| | | Follow-up<br>or ET | | DDMONYYYY<br>HH:MM | Yes | Normal | XX | xxx | XX | XX | xxx/N |

-----

Note: CFB: Change from baseline; NU: Not Useable; CS = Abnormal, Clinically Significant; NCS = Abnormal, Not Clinically Significant; VR = Ventricular Rate; PR=Pulse Rate.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.10.2.S/M ECG: Abnormal Results – Listing (SAD/MAD) Safety Population

| Cohort/Treatment | Subject | Day | Time Point | Date and Time of ECG | ECG Abnormality | Clinically<br>Significant |
|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | Day 1 | Pre-dose | DDMONYYYY<br>HH:MM | Sinus bradycardia otherwise normal ECG, physician comments transcribed as per monitor's request | No |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

#### Listing 16.2.11.S/M Mini-Mental State Examination (SAD/MAD) Safety Population

| Cohort/Treatment | Subject | Day | Date and Time | Score | Results |
|------------------|---------|-----------|-----------------|-------|---------|
| 1/Placebo | XXXX | Screening | DDMONYYYY HH:MM | XX | Normal |

Note: MMSE - Mini-Mental State Examination



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.12.S/M Medical History (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | MH# | Body System/<br>Preferred Term | Condition | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | X | Xxxx/Xxxxx | Xxxxxx | DDMONYY<br>YY | DDMONYYYY | No |

. . .



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.13.S/M Clinical Events (SAD/MAD) Safety Population

| Cohort/<br>Treatment/ | Subject | Clinical Event | Planned time point | Start Date and Time | End Date and Time | Ongoing? |
|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | XXXXXX | Pre-dose | DDMONYYYY | DDMONYYYY | No |
| | | XXXXXX | 5 min | DDMONYYYY | | Yes |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

### Listing 16.2.14.S/M Prior and Concomitant Medications (SAD/MAD) Safety Population

| Cohort/<br>Treatment | Subject | Medication<br># | Drug<br>Class/<br>Preferred<br>Term/<br>Verbatim<br>Term | Medication<br>Information* | Start Date/Stop<br>Date | Ongoing? | Indication | Administered for AE? | Administered for MH? |
|---|---|---|---|---|---|---|---|---|---|
| 1/Placebo | xxxx | 1 | xxxx | xxx/ mg/<br>Once/ Oral | DDMONYYYY/<br>DDMONYYYY | No | Headache | Yes (AE # 4) | No |
| | | 2 | xxxx | xxx/ mg/<br>Once/ Oral | DDMONYYYY | Yes | Xxxxx | No | Yes (MH #2) |
| ••• | | | | | | | | | |

<sup>\*</sup>Dose/Unit/Frequency/Route



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

## Listing 16.2.15.M Electroencephalogram at Screening (MAD) Safety Population

| Cohort/<br>Treatment | Subject | EEG Test Date and Time | Results | Clinically Significant |
|---|---|---|---|---|
| 1/Placebo | xxxx | DDMONYYYY HH:MM | Abnormal | No |



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Figure 14.4.1.S/M – Mean Plasma RP3128 Concentrations – Linear Scale (SAD/MAD)

Safety Population



Programming Notes: Replace XX with corresponding dose of indicated cohort.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

Figure 14.4.2.S/M – Mean Plasma RP3128 Concentrations – Semi-logarithmic Scale (SAD/MAD)

PK Population



Programming Notes: Replace XX with corresponding dose of indicated cohort.



Sponsor: Rhizen Pharmaceuticals SA

Study: Study 15-MR-001

# Figure 14.4.3.X.S/M–Individual Plasma RP3128 Concentrations – Linear Scale (SAD/MAD) (ZZ mg) Safety Population

Programming Notes: Similar to 14.4.1 except graphs will represent individual subject graphs within each cohort. Increase value of X by 1 with each cohort. Replace ZZ with corresponding dose of indicated cohort.

Figure 14.4.X.S/M–Individual Plasma RP3128 Concentrations – Semi-logarithmic Scale (SAD/MAD)

(ZZ mg)

Safety Population

Programming Notes: Similar to 14.4.2 except graphs will represent individual subject graphs within each cohort. Increase value of X by 1 with each cohort. Replace ZZ with corresponding dose of indicated cohort.